### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for a placebo-controlled, double-blind (sponsor open), randomised, crossover study to assess the efficacy, safety, and tolerability of GSK2798745 in participants with chronic cough |
|---|---|---|
| <b>Compound Number</b> | : | GSK2798745 |
| <b>Effective Date</b> | : | 07-SEP-2018 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 207702
- This RAP is intended to describe the efficacy, safety and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Interim Analysis (IA) and Statistical Analysis Complete (SAC) deliverables.

### **RAP Author(s):**

| Approver | Date | Approval Method |
|--------------------------------------|----------------|-----------------|
| PPD | | |
| Principal Statistician | Not Applicable | Not Applicable |
| (Respiratory, Clinical Statistics) | | |
| PPD | | |
| Senior Director | 29-AUG-2018 | Pharma TMF |
| (Respiratory, Clinical Pharmacology) | | |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Development Manager (CPSSO) | 03-SEP-2018 | Pharma TMF |
| Clinical Development Director (Respiratory TAU) | 29-AUG-2018 | Pharma TMF |
| Project Physician (Respiratory TAU) | 02-SEP-2018 | Pharma TMF |
| Data Manager (CPSSO) | 29-AUG-2018 | Pharma TMF |
| PPD Programming Manager (Respiratory, Clinical Programming) | 29-AUG-2018 | Pharma TMF |
| SERM Director (GCSP) | 07-SEP-2018 | Pharma TMF |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Director (Respiratory, Clinical Statistics) | 05-SEP-2018 | Pharma TMF |
| Programming Manager (Respiratory, Clinical Programming) | 30-AUG-2018 | Pharma TMF |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | ODUCTIO | ON | 6 |
| 2. | CLIMAN | | KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | | | |
| | | Change | es to the Protocol Defined Statistical Analysis Plan | 0 |
| | 2.2. | | Objective(s) and Endpoint(s) | |
| | 2.3. | | Design | |
| | 2.4. | Statistic | cal Analyses | / |
| 3. | PLAN | NED AN | ALYSES | 9 |
| | 3.1. | | Analyses | |
| | | 3.1.1. | Review of the Interim Analysis Results | |
| | | 3.1.2. | Conditional Probabilities to Support Sample Size Re- | |
| | | | estimations | 12 |
| | 3.2. | Final Ar | nalyses | |
| | | | • | |
| 4. | ANAL | | PULATIONS | |
| | 4.1. | Protoco | ol Deviations | 14 |
| _ | CONC | | TONG FOR DATA ANALYSES AND DATA HANDLING | |
| 5. | | | IONS FOR DATA ANALYSES AND DATA HANDLING | 4.5 |
| | 5.1. | | IS Freatment & Sub-group Display Descriptors | |
| | 5.1.<br>5.2. | | e Definitions | |
| | 5.2.<br>5.3. | | ntre Studies | |
| | 5.3.<br>5.4. | | | |
| | 5.4.<br>5.5. | | lation of Covariates, Other Strata and Subgroups Considerations for Data Analyses and Data Handling | 10 |
| | 5.5. | | ntions | 17 |
| | | 000 | | |
| 6. | STUD | Y POPU | LATION ANALYSES | 18 |
| | 6.1. | Overvie | ew of Planned Study Population Analyses | 18 |
| _ | | | 141.7/050 | 40 |
| 7. | | | IALYSES | |
| | 7.1. | , | / Efficacy Analyses | |
| | | 7.1.1. | | |
| | | 7.1.2. | ······9 = ····· ( · | |
| | | 7.1.3. | Summary Measure | |
| | | 7.1.4. | Population of Interest | |
| | | 7.1.5. | Statistical Analyses / Methods | |
| | 7.2. | Evnlora | 7.1.5.1. Statistical Methodology Specification | |
| | 1.2. | 7.2.1. | Endpoint / Variables | |
| | | 1.4.1. | 7.2.1.1. Total Cough Counts over 24 Hours | |
| | | | 7.2.1.2. Cough Severity and Urge (VAS) | |
| | | | 7.2.1.3. Leicester Cough Questionnaire (LCQ) | |
| | | 7.2.2. | Missing Data Imputation | |
| | | 7.2.3. | Summary Measure | |
| | | 7.2.4. | Population of Interest | |
| | | 7.2.5. | Statistical Analyses / Methods | |
| | | | 7.2.5.1. Statistical Methodology Specification | |

| 8. | SAFE | ΓΥ ANALY | /SES | 30 |
|---|---|---|---|---|
| | 8.1. | | Events Analyses | |
| | 8.2. | | aboratory Analyses | |
| | 8.3. | Other Sa | fety Analyses | 30 |
| 9. | PHAR | MACOKIN | NETIC ANALYSES | 31 |
| | 9.1. | Primary I | Pharmacokinetic Analyses | 31 |
| | | 9.1.1. | Endpoint / Variables | |
| | | | 9.1.1.1. Drug Concentration Measures | |
| | | | 9.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 9.1.2. | Population of Interest | |
| | | 9.1.3. | Statistical Analyses / Methods | |
| | 9.2. | | ry Pharmacokinetic Analyses | |
| | | 9.2.1. | Endpoint / Variables | |
| | | | 9.2.1.1. Drug Concentration Measures | |
| | | | 9.2.1.2. Derived Pharmacokinetic Parameters | |
| | | 9.2.2. | Population of Interest | |
| | | 9.2.3. | Statistical Analyses / Methods | 32 |
| 10 | POPU | I ATION F | PHARMACOKINETIC (POPPK) AND | |
| 10. | | | NAMIC ANALYSES | 33 |
| | 10.1. | | al Analyses / Methods | |
| 11. | REFE | RENCES. | | 34 |
| 12 | ۸ DDEI | VIDICES | | 35 |
| 12. | 12.1. | | x 1: Protocol Deviation Management and Definitions for Per | 30 |
| | 12.1. | Protocol | Population | 35 |
| | 12.2. | | x 2: Schedule of Activities | |
| | 12.2. | | Protocol Defined Schedule of Events | |
| | 12.3. | | x 3: Study Phases and Treatment Emergent Adverse | |
| | | | | 40 |
| | | | Study Phases and Treatment Emergent Rules for AEs | |
| | | | 12.3.1.1. Study Phases for Concomitant Medication | |
| | 12.4. | Appendix | x 4: Data Display Standards & Handling Conventions | |
| | | | Reporting Process | |
| | | 12.4.2. | Reporting Standards | |
| | | 12.4.3. | Reporting Standards for Pharmacokinetic Data | |
| | 12.5. | Appendix | x 5: Derived and Transformed Data | |
| | | 12.5.1. | General | |
| | | 12.5.2. | Study Population | |
| | | 12.5.3. | Efficacy | |
| | | | 12.5.3.1. Cough Count SI and A&R Dataset | |
| | | | Specifications | |
| | | | 12.5.3.2. Cough Count Missing Data Period Algorithms | |
| | | | 12.5.3.3. Cough Count Imputation Derivations | 54 |
| | | 12.5.4. | Pharmacokinetic | |
| | | 12.5.5. | Population Pharmacokinetic (PopPK) | 54 |
| | | 12.5.6. | Operating Characteristics of Decision Criteria Based on | |
| | | | Conditional Probabilities | |
| | 12.6. | | x 6: Reporting Standards for Missing Data | |
| | | 12.6.1. | Premature Withdrawals | 58 |

| | 12.6.2. | Handling of Missing Data | 58 |
|--------|----------|--------------------------------------------------|-----|
| | | 12.6.2.1. Handling of Missing and Partial Dates | 58 |
| 12.7. | Appendix | 7: Values of Potential Clinical Importance | 59 |
| | 12.7.1. | Laboratory Values | 59 |
| | 12.7.2. | ECG | 60 |
| | 12.7.3. | Vital Signs | 60 |
| 12.8. | Appendix | k 8: Population Pharmacokinetic (PopPK) Analyses | 61 |
| | 12.8.1. | Population Pharmacokinetic (PopPK) Methodology | 61 |
| | | 12.8.1.1. Software | 61 |
| | | 12.8.1.2. Outline | 61 |
| | 12.8.2. | Population Pharmacokinetic (PopPK) Dataset | |
| | | Specification | |
| | | 12.8.2.1. Data Specification | |
| | | 12.8.2.2. Dataset Variable Conventions | |
| 12.9. | | x 9: Pharmacokinetic / Pharmacodynamic Analyses | |
| | 12.9.1. | Pharmacokinetic / Pharmacodynamic Methodology | |
| | | 12.9.1.1. Exposure-Response Relationship | 65 |
| | 12.9.2. | Pharmacokinetic / Pharmacodynamic Dataset | |
| | | Specification | 65 |
| | | 12.9.2.1. Data Specification | |
| | | 12.9.2.2. Dataset Variable Conventions | |
| 12.10. | | x 10: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 12.11. | | x 11: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | | Pharmacokinetic Tables | |
| | | Pharmacokinetic Figures | |
| | | .ICH Listings | |
| 12 12 | | Non-ICH Listings | |
| 1/1/ | ADDEDOIX | C D EXAMOLE MOCK SHELLS TOLD ALA DISDIAVS | 9.5 |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 207702:

| Revision Chronology: | | |
|---|---|---|
| 2017N319286_00 | 31-MAY-2017 | Original |
| 2017N319286_01 | 09-OCT-2017 | Removal of Simplified Nutritional Appetite Questionnaire (SNAQ). |
| 2017N319286_02 | 22-NOV-2017 | Addition of CSSRS at follow-up and updates to emergency unblinding text on request of MHRA. |
| 2017N319286_03 | 25-JUN-2018 | Increasing the upper BMI limit and removing the upper limit for FEV1 |

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 31/MAY/2017), amendment 01 (Dated: 09/OCT/2017), amendment 02 (Dated: 22/NOV/2017) and amendment 03 (Dated: 25/JUN/2018)

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare the efficacy of 7 days dosing<br>of GSK2798745 with placebo in<br>participants with idiopathic or treatment<br>resistant chronic cough | <ul> <li>Total cough counts during day-time hours<br/>following 7 days of dosing</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To compare the safety of GSK2798745<br>with placebo in participants with idiopathic<br>or treatment-resistant chronic cough | <ul> <li>Adverse events (AE), clinical laboratory<br/>values, vital signs, electrocardiogram (ECG),<br/>and other safety biomarkers</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To compare the efficacy of 7 days dosing<br>of GSK2798745 with placebo in<br>participants with idiopathic or treatment<br>resistant chronic cough | <ul> <li>Total cough counts over 24 hours following 7 days of dosing</li> </ul> |
| To compare the efficacy of 7 days dosing<br>of GSK2798745 with placebo at<br>improving patient reported outcomes in<br>participants with idiopathic or treatment-<br>resistant chronic cough | <ul> <li>Change from baseline cough severity and urge to cough visual analogue scale (VAS)</li> <li>Change from baseline Leicester Cough Questionnaire (LCQ) score</li> </ul> |
| To evaluate the pharmacokinetics (PK) of<br>GSK2798745 and its M1 metabolite in<br>participants with idiopathic or treatment<br>resistant chronic cough | <ul> <li>Plasma concentrations of GSK2798745 and<br/>derived PK parameters, as data permit</li> </ul> |

## 2.3. Study Design



# 2.4. Statistical Analyses

The study is designed to estimate the effect of GSK2798745 relative to placebo on day-time cough counts following seven days of dosing. Day-time cough count totals will be

derived from the total number of coughs during the first 10 hours following dosing, during which the participant is expected to be awake.

The inference to be carried out will be with respect to the following hypothesis:

• Treatment with GSK2798745 leads to a reduction in day-time 10-hour cough count totals compared with placebo.

The above hypothesis will be investigated in this study by means of a Bayesian approach, which will assume a non-informative prior distribution. It is anticipated that the day-time 10-hour cough count totals will be log-transformed before statistical analysis, and hence the treatment effect will be evaluated in terms of a ratio of day-time cough count totals (GSK2798745 / placebo), with corresponding 90% credible interval. A day-time cough count total of at least 30% less for GSK2798745 than for placebo is of interest. The posterior probability that the true ratio is less than 0.7 will be obtained and will be referred to as PP (ratio<0.7).

### 3. PLANNED ANALYSES

# 3.1. Interim Analyses

An interim analysis is planned after at least 12 participants have completed both dosing periods and will be based on day-time 10h total cough count data, as well as supporting PK data, if required. PK data will remain blinded if assessed as part of any interim analyses.

An ongoing review will take place to ensure that compliance to study drug and validity of cough data are acceptable for the interim analysis. For cough data to be valid, at least 60% of the recording time during the first 10 hours must be available, See Section 7.1.2. If compliance or cough data are deemed to be invalid for the first 12 participants who have completed both dosing periods, then consideration will be given to waiting for additional participants to meet the minimum of 12 participants with valid data for analysis.

The primary objectives of the interim analysis are to:

- i) Stop the study on the grounds of futility
- ii) Re-estimate the sample size based on the treatment effect and variability observed at the time of the interim.

As the study is double blind (sponsor-open), the results will be made available to a core subset of the GSK study team, who will review the data (treatment level only), before making a decision on whether to stop the study for futility or adjust the sample size. Decisions from the interim analyses and details of members of the GSK study team who reviewed the results, will be documented in the interim results meeting minutes. Any adjustment to the sample size will be communicated to the sites.

The sample size re-estimation will be supplemented by deriving conditional probabilities. As a result of this supportive information, the sample size could be revised either upwards or downwards from the planned sample size of 24 evaluable participants, but the target number of evaluable participants will not exceed 40 participants.

The interim analysis will be performed by GSK Clinical Statistics and only the responsible statistician(s) (including QC statistician(s)) and programmers will have access to the study reporting area where the individual participant data which will be unblinded for the interim analyses. Unblinded treatment sequences will only be made available for participants who will be included in the interim analysis. A list of randomisation numbers of those who have completed the relevant treatment periods for the interim analysis will need to be provided by the study manager or designee, to release the treatment sequence codes.

The interim analysis will use clean efficacy data (cough count data provided by Vitalograph and subject to QC and cleaning processes) and will be supplemented by the following in stream data from the eCRF for use in standard HARP programs; cough dates and times, exposure and compliance information, demography data and stratification responses. SI datasets for the specified eCRF data will be provided by Data Management

to a level as clean as possible at the time of the interim, with data as complete as possible (up to Period 2 Day 8) for the randomised participants who will be included in the interim analysis. Statistics and programming will cut the data (subset) based on the list of randomised participants available for the interim analysis.

It is expected that outputs from the Interim Analysis will not be required for the Clinical Pharmacology Study Report (CPSR) as only final data will be formally reported. The CPSR will provide brief details that an interim analysis was performed and sample size subsequently increased or decreased.

Details for the statistical analysis of total 10h day-time cough counts are provided in Section 7.1.5. The proposed outputs to be provided for the interim analysis are as follows, refer to Section 12.11 for further details and examples:

- Summary of statistical analysis (including treatment ratio and 90% credible intervals along with posterior probabilities of interest, see example EF\_T1). A preliminary assessment of carry-over and/or period by treatment interaction will be investigated as part of this analysis. The analysis will be based on imputed 10h totals (see Section 7.1.2).
- Figure of treatment group geometric means and 95% CIs for both baseline and Day 7 10h day-time cough counts (see example EF\_F1)
- Figure as above split by treatment period to assist with assessment of carryover and/or period by treatment interaction
- Figure of overall hourly profiles (0-10h), geometric (or arithmetic dependent on data) means ± 95% CIs for GSK2798745 vs Placebo at each hourly timepoint (see example EF F2).

#### 3.1.1. Review of the Interim Analysis Results

Once the interim results are available, the following steps will be taken to support decision making moving forward.

#### 1. Assessment of results

The results from the interim analysis (as well as final analysis) will be compared with pre-defined criteria for a positive and negative study as follows:

The pre-defined criterion for a **positive study** is a posterior probability of more than 70% that the true treatment ratio (GSK2798745 / placebo) is less than 0.7, i.e. PP(ratio<0.7)>70%.

The pre-defined criterion for a <u>negative study</u> is a posterior probability of less than 30% that the true treatment ratio (GSK2798745 / placebo) is less than 0.7, i.e. PP(ratio<0.7)<30%.

There is a grey area in which neither criterion is satisfied.

## 2. Sample Size Re-estimation

A graphic will be produced displaying the conditional probability of achieving various sample sizes (see Section 3.1.2) under positive and negative scenarios. From these estimates, an initial re-estimated sample size will be identified.

#### 3. Supportive Information

Further information to be considered, which may influence what the final sample size will be:

- The change in conditional probability achieved vs. the change in the number of participants required to achieve it, e.g. increasing the sample size by 10 participants to achieve an extra 2% of conditional probability might not be deemed worthwhile
- The results of the Bayesian mixed model analysis of the interim data, i.e. the treatment ratio and variability observed in the interim data, and the probabilities that the true treatment ratio is less than 0.5, 0.7 and 1 based on the interim data
- Information on the profile of coughing over time as provided by the figure of geometric means and 95% CI for cough counts at each hourly interval
- Results of any further exploratory analyses of the cough count data dependent on the interim analysis results

#### 4. Final Sample Size Decision

The estimate of sample size in the protocol is 24. The maximum revised sample size can be up to 40 evaluable participants (maximum 48 randomised). Factors as described in #1, #2 and #3 above will be reviewed to support a decision on increasing or decreasing the sample size from the planned 24 participants.

Based on the results of the interim analyses, if there is strong evidence of a **positive** outcome based on conditional probabilities then this may, once other factors as described above have been considered, lead to a reduction in sample size equal to **the total number of participants who have completed the study together with those who are currently in the study**.

If there is strong evidence of a **negative** outcome based on conditional probabilities and there are no further factors which suggest that more information is needed, then the sample size may be reduced, again to equal **the total number of participants who have completed the study together with those who are currently in the study.** 

In both cases, the total sample size will be estimated closer to the interim based on recruitment at the time and all ongoing participants will complete the study. Strong evidence would include results from the interim that meet our pre-defined criteria and the supporting conditional probabilities indicating a reduction in sample size to close to the interim N.

The full rationale for the decision on the final sample size, incorporating any considerations beyond the primary conditional probabilities, will be documented in the interim analysis meeting minutes.

# 3.1.2. Conditional Probabilities to Support Sample Size Re-estimations

Sample size re-estimation will be supported by conditional probabilities of meeting the pre-defined positive and negative criteria for the study. This method utilises the data we have from the interim, but makes assumptions on the future data based on different scenarios. When calculating conditional probabilities, scenarios as detailed below will be considered.

The sample size giving a 90% conditional probability of meeting the **positive** criterion at the end of the study, based on the variability observed in the <u>interim sample</u> and based on the variability <u>assumed for the protocol</u>, conditioning on:

- o a treatment ratio of 0.5 for the post-interim data
- o the treatment ratio observed in the interim sample for the post-interim data

The sample size giving approximately 90% conditional probability of meeting the <u>negative</u> criterion at the end of the study, based on the variability observed in the interim sample and based on the variability assumed for the protocol, conditioning using:

- o a treatment ratio of 0.95 for the post-interim data
- o the treatment ratio observed in the interim sample for the post-interim data

All scenarios will be evaluated as part of the interim results review, however, the positive and negative study scenarios that utilise the interim observed variability and condition on the treatment ratio observed in the interim sample would be the key focus for decision making (yellow and brown dotted lines in the example graphic below).

#### **Example of Graphic to illustrate Conditional Probabilities at the Interim**

The graphic below shows an example of a 'conditional probabilities' graphic. In this example, it is based on overwhelming success at the interim, a ratio of 0.45 observed. If we assume that effect continues in the study (i.e., yellow line, conditioning on the interim ratio of 0.45) then there is no impact on the probability of meeting the success rule as the sample size increases, this is maintained at  $\sim 100\%$  as we have already reached our success criteria. In this instance, we may continue the study until the currently randomised participants could complete the study, without randomising further participants.

Similarly, there is no impact on the probability of meeting the negative rule, brown dotted line, conditioning on the interim ratio of 0.45. This stays at  $\sim$ 0% (again as we have already met the success criteria).

The green line shows the impact of observing a very good drug effect at the interim but the probability of declaring a negative study if we still believe our true effect may be 'no/little effect', i.e. conditioning on a ratio of 0.95. In this case, we would have  $\sim 25\%$ 

probability of declaring a negative study with N=24 patients if we continued this study, when the true effect was in fact 'no effect'.

For the current study, if at the interim we have observed a good effect (ratio close to 0.70) then this graphic will help determine the sample size to continue with based on the variability observed at the interim. If the interim variability is lower than originally predicted, as defined in the protocol, then we may meet our success criteria at that point with a ratio of 0.7 or less. If the variability is as expected or higher, we may need to continue the study to reach our success probability and this graphic will guide us to the sample size most likely to achieve success.



Example Study Conditional Probabilities Across a Range of Final Sample Sizes Success Rule = Pr(Treatment Ratio<0.7)>0.70, Negative Rule = Pr(Treatment Ratio<0.7)<0.30 SigmasqW=0.280 (SDwmult=100)

Example operating characteristics for the above scenarios are presented in Section 12.5.6.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol (and subject to decisions made based on the interim analyses).
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met. Note that the study is being run as sponsor open, however for the interim analyses, only a partial randomisation schedule will be made available to GSK Clinical Statistics, applicable

to those participants who completed two dosing periods and for whom cough data will be transferred.

4. Randomisation codes have been distributed according to RandAll NG procedures.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants screened and for whom a record exists on the study database | Disposition (including reasons for screening failures) |
| All Subjects | All randomized participants who take at least 1 dose of study treatment. Participants will be analysed according to the treatment they actually received | <ul><li>Study Population</li><li>Efficacy</li><li>Safety</li></ul> |
| Pharmacokinetic<br>(PK) | All randomized participants who take at least 1 dose of study treatment and for whom a pharmacokinetic sample <sup>a</sup> was obtained and analysed | • PK |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the current version of the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the eligibility page of the eCRF.

<sup>&</sup>lt;sup>a</sup> refers to sample taken for the analysis of GSK2798745 and metabolite OR sample taken for analysis of Atorvastatin.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Note that all displays (Tables, Figures & Listings) will use the term 'Subjects'.

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description | Order in TLF |
| Α | Placebo | Placebo | 1 |
| В | GSK2798745 | GSK2798745 | 2 |

Treatment comparisons will be displayed as follows using the descriptors as specified: GSK2798745 vs Placebo

### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. Baseline definitions are applicable to <u>each period</u>.

| Parameter | Study Asses | Baseline Used in | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Efficacy | | | | |
| Total day-time cough count | | Х | | Day -1 |
| Total 24 hour cough count | | Х | | Day -1 |
| Cough Severity (VAS) | Х | Х | | Day -1 |
| Urge to Cough (VAS) | | Х | | Day -1 |
| Leicester Cough<br>Questionnaire (LCQ) | | Х | | Day -1 |
| Columbia Suicidality<br>Severity Rating Scale<br>(CSSRS) | Х | Х | | Day -1 |
| Safety | | | | |
| Labs | Χ | | Xa | Day 1 (Pre-Dose) |
| ECGs | Xp | | X | Day 1 (Pre-Dose) |
| Vital Signs | Xp | | X | Day 1 (Pre-Dose) |
| Audiometry | | Χ | | Day -1 |

<sup>&</sup>lt;sup>a</sup> Can be completed on Day 1 (pre-dose) or Day -1

Unless otherwise stated, if baseline data is missing no derivation (e.g., change from baseline) will be performed and baseline will be set to missing.

For statistical analyses (for example, Bayesian mixed model) in a crossover design the following baseline derivations may apply:

- Baseline is defined as the 10h daytime cough count total observed pre-dose (Day -1) of each treatment period. This can also be referred to as 'period-specific baseline'.
- **Subject-level baseline** is defined as the mean of the two period-specific baseline readings (the Day -1 10h cough count total from each of the two treatment periods) for each participant.
- **Period-level baseline** (or 'adjusted period-specific baseline') is defined as the difference between the baseline ('period-specific baseline') and 'subject-level baseline' for each period and each participant (i.e., the 'period-specific baseline' minus 'subject-level baseline' in each period).

The statistical modelling may include terms for 'subject-level baseline' and 'adjusted period-specific baseline'.

#### 5.3. Multicentre Studies

In this multicentre study (UK), enrolment will be presented by investigative site in listings. Data will be summarised for all sites combined. A treatment-by-centre interaction may be investigated in the statistical analysis if sufficient data is available.

# 5.4. Examination of Covariates, Other Strata and Subgroups

The list of covariates, strata and subgroups may be used in descriptive summaries and statistical analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|---|---|
| Strata | <b>Prior cough study stratification</b> : Participants who did/did not take part in previous cough studies in the last 12 months. This is a stratification factor within the randomisation and will also be included in the database. The effect of this will be investigated as part of the statistical analysis. |
| Covariates | <b>Centre</b> If sufficient data is available, the effect of centre on the primary endpoint will be investigated. For data displays, data from centres will be combined unless otherwise specified in the list of outputs. |
| Subgroups | No subgroups are pre-specified, will be considered on an adhoc basis if required. |

<sup>&</sup>lt;sup>b</sup> Performed in triplicate

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 12.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 12.4 | Appendix 5: Derived and Transformed Data |
| 12.6 | Appendix 6: Reporting Standards for Missing Data |
| 12.7 | Appendix 7: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the All Subjects population, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 11: List of Data Displays.

#### 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

#### 7.1.1. Endpoint / Variables

The primary efficacy endpoint is the total day-time cough count (10 hours).

This will be calculated from the time of the monitor being attached i.e., immediately after dosing on Day 7 to 10h past the start time of monitoring. The participant is expected to be awake during this period.

In addition, hourly total cough counts will be calculated for descriptive purposes. These will be measured in 60 minute intervals post the start time of the device monitoring.

A dataset of cough events (one row per cough) will be provided by Vitalograph. Four 24 hour sessions of data are expected for each participant (Period 1 Day -1, Period 1 Day 7, Period 2 Day -1 and Period 2 Day 7). This data will be made available to S&P via Data Management. Vitalograph will also provide an additional file (SAS format) containing information related to each session with regards to removal and re-attachment of the cough monitor as well as clearly defined sleep periods within each session. Further details on the cough count data to be transferred is provided in a Cough Analysis Plan written by Vitalograph.

Further details of the file structure for the cough count totals and additional session information are provided in Section 12.5.3.

## 7.1.2. Missing Data Imputation (0-10h)

In the unlikely event that a participant removes the cough monitor, turns off the device, has a period of data that cannot be analysed (flagged area) or other reasons for potential missing cough monitoring during the 10h from the start of the monitoring period, then the participant's cough profiles will be assessed to determine whether it is best to pro-rata the results based on the full 10h period, or to calculate the day-time 10h cough count total as missing. Should any data be pro-rated the resulting number of coughs will be rounded to the nearest integer value. As a rule of thumb, allowance for pro-rated data can be made if at least 60% of the first 10 hours of monitoring includes valid cough monitoring data (e.g., the monitor is attached and working for at least 6 out of the first 10 hours).

For example, if a participant recorded 200 coughs between 0 and 8 hours but the monitor was removed for the next 2 hours, we could estimate the 2 hour cough count as 50, with a resulting imputed 10h total of 250 coughs.

Pro-rated missing data rules as above will also be applied separately to <u>hourly cough</u> count totals, where at least 60% of the hourly interval has valid cough monitoring recorded.

Note that the rules applied to hourly intervals vs the 10h total, could result in the sum of the imputed hourly interval cough totals not being equal to the 10h total. For example, if a participant had an error with the device during the first hour resulting in no cough data then this hourly interval could not be imputed (as > 60% missing). However, if further monitoring was complete then the 10h total could use data from the remaining 9 hours to impute a cough count for the first hour. Hence in this example, the 10h total would be slightly higher than the sum of individual hourly totals.

Information regarding removal and re-attachment, late attachment, early termination/stoppage, sleep periods and flagged periods during the cough monitoring will be provided by Vitalograph in a separate information file (see Section 7.1.1). Dates and times of the events within this file will be merged with the databased cough data to assess the extent of missing time periods. Sleep periods will also be identified and will be classed as missing data, if the sleep period is within the first 10 hours of monitoring.

Further details of the file structure for the cough count totals and additional session information, plus further examples of missing data imputation and associated algorithms are provided in Section 12.5.3.

Details of any imputation will be fully documented and highlighted in participant listings.

### 7.1.3. Summary Measure

The summary measure for the primary analysis is the adjusted median posterior difference and 90% credible interval for GSK2798745 vs Placebo at Day 7 for total day-time cough counts (10 hours). A log-transformation of the cough count data is expected prior to analysis, in which case, the treatment effect will be evaluated in terms of a ratio of total day-time cough counts (GSK2798745/Placebo).

The primary analysis will be performed on pro-rated/imputed 10h cough count totals.

A sensitivity analysis will be conducted for the final analysis based on raw unimputed data.

### 7.1.4. Population of Interest

The primary efficacy analyses will be based on the All Subjects population, unless otherwise specified.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Total day-time cough counts (10 hours)

## **Model Specification**

- The description below describes the current thinking of how to analyse these endpoints. The
  proposed model will be assessed, and if not appropriate alternative models could be used.
- The data will be inspected prior to analysis to determine whether a data transformation is required. A log-transformation is expected for the total cough count data. Any data transformations will be applied to observed individual daytime 10h total cough counts prior to any modeling or derivations (e.g. prior to deriving subject baseline or period-adjusted baseline)
- A Bayesian mixed effects model (fitted using SAS PROC MCMC), will be used to model the total day-time cough counts (10 hours) after 7 days of dosing.
- Covariates for period, treatment, centre and previous cough study participation (stratification factor in the randomisation) will be included as fixed effects. Adjusted period-specific baseline and subject-level baseline will be included as continuous parameters. Subject will be included as a random effect. A treatment by period interaction will be included to investigate preliminary carry-over effects and/or a period by treatment interaction and if deemed appropriate an analysis by period may be performed. The assessment of the interaction will be performed using the equivalent PROC MIXED model and graphical representation.
- An unstructured variance-covariance matrix will be fitted. A non-informative prior distribution will be assumed for posterior probabilities.
- Examination of additional covariates (for example Age group) may take place, if data permit.
   In this case, the equivalent model may be fitted in PROC MIXED and the covariate assessed at a 10% alpha level. The final Bayesian model would then be fitted based upon the final model (after covariate examination) obtained using PROC MIXED.
- Appropriate combinations of the model parameters will be used to obtain the posterior distribution for the GSK2798745 vs placebo on Day 7. Total 10h day-time cough counts will be represented via adjusted posterior medians for GSK2798745 and placebo, as well as associated 95% equi-tailed credible intervals. These results will be presented within tabular and graphical form after data has been back transformed.
- The difference in total day-time cough counts between GSK2798745 and placebo, will be represented via an adjusted median, as well as associated 90% equi-tailed credible interval. These results will be presented within tabular form after data has been back transformed, hence representing the ratio of GSK2798745/placebo.
- The posterior distributions will also be used to produce several posterior probability statements, presented in tabular format; the most important being the probability that the true ratio (GSK2798745/placebo) is less than 0.7, representing a 30% reduction in total day-time cough counts on GSK2798745. Probabilities that the true ratio is less than 1 (any effect) and less than 0.5 (excellent effect) will also be constructed.

## **Model Checking & Diagnostics**

- Fixed effects will be assigned a non-informative prior of N(0, Var=1E6) and may be entered as separate univariate priors or as part of a multivariate distribution (variance covariance structure with zeros for off diagonals) in model hyperpriors.
- The non-informative UN priors should be an inverse Wishart distribution. If the equivalent of

an unstructured variance covariance matrix does not fit then an AR(1) w/Random Effect structure may be considered, with non-informative priors  $\phi$ ~U[-1,1] for the off diagonal elements and  $\sigma$ <sup>2</sup> ~ invGamma(0.0001, scale=0.0001). Example, for N=2:

$$UN = \begin{pmatrix} \sigma_1^2 & \sigma_{21} \\ \sigma_{21} & \sigma_2^2 \end{pmatrix}$$

$$AR(1) = \begin{pmatrix} 1 & \varphi \\ \varphi & 1 \end{pmatrix} * \sigma^2$$

•

- Centring of any continuous covariates will take place at the input dataset stage: (valuei average) for each subject i.
- Examination of trace plots to assess convergence. Autocorrelation plots and lag summary table to assess the degree of autocorrelation. Monte Carlo standard errors compared to posterior standard deviations (target would be MCSE/SD<0.01).</li>
- Number of burn ins, thinning, starting points, number of posterior draws to take (10,000 may be
  a suitable starting default) will be customised to each model and may not be possible to specify
  in advance but will be modified to ensure satisfactory diagnostics are produced.
- For robustness, where non-informative priors are used the equivalent PROC MIXED model
  may be fitted (no output from this would be reported) and LS Means and estimates of
  treatment differences/ratios compared to the results obtained from the PROC MCMC analysis.
- Model assumptions will be applied, but appropriate adjustments may be made based on the data. A log-transformation is expected to total day-time 10h cough counts.

#### **Model Results Presentation**

- Summary table for total 10h day-time cough counts
- Listing of total hourly cough counts and 10h day-time cough counts by timepoint (baseline and Day 7) and treatment
- Individual hourly subject profiles (4 subjects per page) of day-time cough counts by treatment group and timepoint (0-10h)
- Boxplots of cough counts by treatment group and hourly timepoint (0-10h)
- (A) (\*) Figure of geometric means  $\pm$  95% CIs of cough counts by treatment group and hourly timepoint (0-10h) (data permitting, arithmetic means may be presented)
- (B) (\*) Figure of geometric means ±
- 95% Cls by treatment for Day -1 vs Day 7 10h day-time cough count totals
- Figure of subject by total 10h day-time cough counts and treatment
- Figure of individual changes from baseline for 10h cough counts (Day -1) to Day 7 by treatment group
- (\*) Summary table of statistical analysis of total 10h day-time cough counts including: adjusted posterior medians and 95% credible intervals by treatment, estimated posterior median treatment effect (ratio GSK2798745/placebo) and 90% credible interval, posterior probabilities of interest (ratio<1, ratio<0.7 and ratio<0.5) based on imputed data
- Summary table of statistical analysis of total 10h day-time cough counts including: adjusted
  posterior medians and 95% credible intervals by treatment, estimated posterior median
  treatment effect (ratio GSK2798745/placebo) and 90% credible interval, posterior probabilities
  of interest (ratio<1, ratio<0.7 and ratio<0.5) sensitivity analysis not accounting for missing</li>

data

- Figure of statistical analysis adjusted medians and 95% credible intervals by treatment group
- Figures (A) and (B) above may also be reproduced split by stratification factor (prior study participation)
- (\*) To be produced for the interim analysis

#### Sensitivity and Supportive Analyses

- Period 1 analysis: Should the interim analysis or final analysis provide evidence of a possible carryover effect from the treatment of GSK2798745 from period 1 into period 2 and/or period by treatment interaction, then an analysis of period 1 data only may take place.
- In this case, a Bayesian model will be fitted including terms for treatment, stratification factor, centre and period 1 baseline. An equivalent PROC MIXED model will be fitted for robustness or as an alternative method. Adjusted posterior medians will be provided as described previously.

## 7.2. Exploratory Efficacy Analyses

## 7.2.1. Endpoint / Variables

#### 7.2.1.1. Total Cough Counts over 24 Hours

The endpoint is total cough counts over 24 hours. This will be calculated from the time of the monitor being attached i.e., immediately after dosing on Day 7 to 24h past the start time of monitoring.

In addition, hourly total cough counts will be calculated for descriptive purposes. These will be measured in 60 minute intervals post the start time of the device monitoring.

#### 7.2.1.2. Cough Severity and Urge (VAS)

The endpoints are:

- Change from baseline in cough severity
- Change from baseline in urge to cough

Both will be measured on a 0-100mm visual analogue scale, where 0 represents a good response (no severity or urge to cough) and 100 represents a poor response (extremely severe cough or severe urge to cough).

#### 7.2.1.3. Leicester Cough Questionnaire (LCQ)

The endpoint is change from baseline in Leicester Cough Questionnaire total and domain scores (LCQ).

The Leicester Cough Questionnaire consists of 19 questions, each with a 7 point Likert response scale., where 1 represents a poor response (affecting quality of life) and 7 represents a good response. The 19 questions fall into 3 domains as follows:

Physical: 1, 2, 3, 9, 10, 11, 14, 15

Psychological: 4, 5, 6, 12, 13, 16, 17

Social: 7, 8, 18, 19

For each of the above domains, the domain score will be calculated as the sum of the scores for the questions in that domain, divided by the number of items in the domain. The LCQ Total Score is then calculated as the sum of the three domain scores, and ranges from 3 to 21. A higher score indicates a better health status.

## 7.2.2. Missing Data Imputation

## **Total cough counts 24h**

Please refer to Section 7.1.2 detailing that at least 60% of cough monitoring data must be available. The 60% cut-off will apply to data over 24 hours, but will apply to intervals within the 24 hours as detailed below. The totals from these intervals will be summed to provide a 24 hour total.

Two methods of determining intervals within the 24h will be used:

- 1. Where only one sleep period is recorded (will be for the majority of participants), then the 24h data will be split into 'awake' and 'asleep' intervals as determined by the sleep start/stop times provided by Vitalograph. Within each 'awake' and 'asleep' interval if at least 60% of the monitoring data is available, then missing data will be imputed from the remaining data within that interval.
- 2. If there is more than one sleep period, or where there is no information on sleep times, then the 24 hour data will be split into three distinct intervals: 0-12h (12h) representing an awake period, 12-20h (8h) representing most likely sleep interval and 20-24h (4h) representing the last 4 hours of monitoring on the second day of wearing the device (morning). Missing data, based on the 60% rule, will then be imputed within each of these intervals.

Each interval as described above will be assessed against the 60% criteria. However, in the event that one or more intervals cannot be imputed (as less than 60% of data is available), the following will apply:

- If the overall amount of data available over the 24h period is still at least 60%, then an individual interval can be imputed (regardless of 60% rule within that interval), provided the monitor was switched on and recording for some part of the interval of interest.
- If an interval is completely missing, but the full 24h period still has at least 60% of data, then the imputed 24h total will be calculated based on the full 24h period of data available, ignoring sleep/awake intervals.

If there is no missing data, then the imputed variable will be set to the raw cough total. If there is less than 60% of data available over the 24h period then the imputed variable will be set to missing.

Pro-rated missing data rules as above will also be applied separately to <u>hourly cough</u> count totals over the 24h period, where at least 60% of the hourly interval has valid cough monitoring recorded. For hourly intervals, awake and asleep times will not be evaluated.

On review of the data and potential for scenarios outside of those described above, the most appropriate method of imputation will be used. Any changes to the above methods will be described in the CSR.

Details of any imputation will be fully documented and highlighted in participant listings. Please refer to Section 12.5.3 with regards to further details on variable naming and the proposed structure of an A&R dataset for cough counts.

#### **Severity and Urge to Cough (VAS)**

Data will not be imputed.

#### Leicester Cough Questionnaire (LCQ)

Data for the individual responses that contribute to the domain and total scores will not be imputed. Missing data is unlikely as the questionnaires are completed at clinic visits. In the event of a missing individual question, the domain scores will still be calculated, with the number of questions answered modified in the calculation, see Section 7.2.1.3.

### 7.2.3. Summary Measure

The summary measure for total 24h cough counts is the adjusted median posterior difference and 90% credible interval for GSK2798745 vs Placebo at Day 7.

The analysis will be performed on pro-rated/imputed 24h cough count totals and a sensitivity analysis will be conducted for the final analysis based on raw unimputed data.

The summary measure for change from baseline in cough severity and urge to cough (VAS) is the adjusted median posterior difference and 90% credible interval for GSK2798745 vs Placebo at Day 7 (pre-dose).

The summary measure for change from baseline in total and domain LCQ scores is the adjusted median posterior difference and 90% credible interval for GSK2798745 vs Placebo at Day 7 (pre-dose).

#### 7.2.4. Population of Interest

The exploratory efficacy analyses will be based on the All Subjects population, unless otherwise specified.

## 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 7.2.5.1. Statistical Methodology Specification

### **Endpoint / Variables**

Total cough counts over 24 hours

#### **Model Specification**

 Data for this endpoint will be analysed in the same way as for the primary endpoint, see Section 7.1.5.1

### **Model Checking & Diagnostics**

Refer to Section 7.1.5.1

#### **Model Results Presentation**

- Summary table for total 24h day-time cough counts
- Listing of total hourly cough counts and 24h day-time cough counts by timepoint (baseline and Day 7) and treatment
- Individual hourly subject profiles (4 subjects per page) of day-time cough counts by treatment group and timepoint (0-24h)
- Boxplots of cough counts by treatment group and hourly timepoint (0-24h)
- (A) Figure of geometric means  $\pm$  95% CIs of cough counts by treatment group and hourly timepoint (0-24h) (data permitting, arithmetic means may be presented)
- (B) Figure of geometric means  $\pm$  95% CIs by treatment for Day -1 vs Day 7 24h cough count totals
- Figure of subject by total 24h cough counts and treatment
- Figure of individual changes from baseline for 24h cough counts (Day -1) to Day 7 by subject and treatment group
- Summary table of statistical analysis of 24h day-time cough counts including: adjusted posterior medians and 95% credible intervals by treatment, estimated posterior median treatment effect (ratio GSK2798745/placebo) and 90% credible interval, posterior probabilities of interest (ratio<1, ratio<0.7 and ratio<0.5) based on imputed data
- Summary table of statistical analysis of 24h day-time cough counts including: adjusted posterior medians and 95% credible intervals by treatment, estimated posterior median treatment effect (ratio GSK2798745/placebo) and 90% credible interval, posterior probabilities of interest (ratio<1, ratio<0.7 and ratio<0.5) sensitivity analysis not accounting for missing data</li>
- Figure of statistical analysis adjusted medians and 95% credible intervals by treatment group
- Figure (A) and Figure (B) above may also be reproduced split by stratification factor (prior study participation)

## Subgroup Analyses

Refer to Section 7.1.5.1

#### **Sensitivity and Supportive Analyses**

Refer to Section 7.1.5.1

#### **Endpoint / Variables**

• Change from baseline to Day 7 (pre-dose) in cough severity and urge to cough (VAS)

#### **Model Specification**

- VAS is measured on a 0 to 100mm scale.
- The description below describes the current thinking of how to analyse these endpoints. The
  proposed model will be assessed, and if not appropriate alternative models could be used.
- The data will be inspected prior to analysis to determine whether a data transformation is required.
- A Bayesian mixed effects model (fitted using SAS PROC MCMC), will be used to model the change from baseline to Day 7 (pre-dose) VAS endpoints as detailed above.
- Covariates for period, treatment, centre and previous cough study participation (stratification factor in the randomisation) will be included as fixed effects. Adjusted period-specific baseline and subject-level baseline will be included as continuous parameters. Subject will be included as a random effect. A treatment by period interaction will be included to investigate preliminary carry-over effects and/or a period by treatment interaction and if deemed appropriate an analysis by period may be performed.
- An unstructured variance-covariance matrix will be fitted. A non-informative prior distribution will be assumed for posterior probabilities.
- Examination of additional covariates (for example Age group) may take place, if data permit.
   In this case, the equivalent model may be fitted in PROC MIXED and the covariate assessed at a 10% alpha level. The final Bayesian model would then be fitted based upon the final model (after covariate examination) obtained using PROC MIXED.
- Appropriate combinations of the model parameters will be used to obtain the posterior distribution for the GSK2798745 vs placebo.
- Change from baseline to Day 7 (pre-dose) VAS endpoints will be represented via adjusted
  posterior medians for GSK2798745 and placebo, as well as associated 95% equi-tailed
  credible intervals. These results will be presented within tabular and graphical form after data
  has been back transformed (if necessary).
- The difference in change from baseline to Day (pre-dose) VAS endpoints between GSK2798745 and placebo, will be represented via an adjusted median, as well as associated 90% equi-tailed credible interval. These results will be presented within tabular form after data has been back transformed to represent a ratio (if necessary).
- The posterior distributions will also be used to produce posterior probability statements, presented in tabular format; for example, the probability that the true difference (GSK2798745-placebo) in change from baseline in VAS is less than 0, less than -17mm or less than -30 mm, i.e. any treatment difference in favour of GSK2798745, a difference of 17 mm in favour of GSK2798745 or a difference of 30 mm in favour of GSK2798745.

## **Model Checking & Diagnostics**

Refer to Section 7.1.5.1

#### **Model Results Presentation**

- Summary table by visit and treatment group (separate outputs for severity and urge)
- Summary table of change from baseline by treatment group (separate outputs for severity and urge)
- Listing of severity and urge to cough VAS by timepoint (baseline and Day 7) and period (endpoints in one listing)
- Figure of absolute mean VAS  $\pm$  95% CI by timepoint and treatment group (separate graphic for severity and urge)
- Summary table of statistical analysis of change from baseline to Day 7 (pre-dose): adjusted posterior medians and 95% credible intervals by treatment, estimated posterior median treatment effect and 90% credible interval, posterior probabilities of interest (difference <0, difference <-17 mm and difference <-30 mm on VAS scale) (separate outputs for severity and urge)</li>
- Figure of statistical analysis adjusted medians and 95% credible intervals by treatment group (separate outputs for severity and urge)

#### Subgroup Analyses

Refer to Section 7.1.5.1

#### **Sensitivity and Supportive Analyses**

Refer to Section 7.1.5.1

#### **Endpoint / Variables**

• Change from baseline to Day 7 (pre-dose) in LCQ domain mean scores and total score

#### **Model Specification**

- LCQ is on a 1 to 7-point scale
- The description below describes the current thinking of how to analyse these endpoints. The proposed model will be assessed, and if not appropriate alternative models could be used.
- The data will be inspected prior to analysis to determine whether a data transformation is required.
- A Bayesian mixed effects model (fitted using SAS PROC MCMC), will be used to model the change from baseline to Day 7 (pre-dose) LCQ endpoints as detailed above.
- Covariates for period, treatment, centre and previous cough study participation (stratification factor in the randomisation) will be included as fixed effects. Adjusted period-specific baseline and subject-level baseline will be included as continuous parameters. Subject will be included as a random effect. A treatment by period interaction will be included to investigate preliminary carry-over effects and/or a period by treatment interaction and if deemed appropriate an analysis by period may be performed.
- An unstructured variance-covariance matrix will be fitted. A non-informative prior distribution will be assumed for posterior probabilities.
- Examination of additional covariates (for example Age group) may take place, if data permit.
   In this case, the equivalent model may be fitted in PROC MIXED and the covariate assessed at a 10% alpha level. The final Bayesian model would then be fitted based upon the final

- model (after covariate examination) obtained using PROC MIXED.
- Appropriate combinations of the model parameters will be used to obtain the posterior distribution for the GSK2798745 vs placebo.
- Change from baseline to Day 7 (pre-dose) LCQ endpoints will be represented via adjusted
  posterior medians for GSK2798745 and placebo, as well as associated 95% equi-tailed
  credible intervals. These results will be presented within tabular and graphical form after data
  has been back transformed (if necessary).
- The difference in change from baseline to Day 7 (pre-dose) LCQ endpoints between GSK2798745 and placebo, will be represented via an adjusted median, as well as associated 90% equi-tailed credible interval. These results will be presented within tabular form after data has been back transformed to represent a ratio (if necessary).
- The posterior distributions will also be used to produce several posterior probability statements, presented in tabular format; the most important being the probability that the true difference (GSK2798745-placebo) is > 0, > 1 and > 1.3, i.e., any treatment difference or a difference of 1 or 1.3 points on the LCQ domain/total score in favour of GSK2798745.

## **Model Checking & Diagnostics**

Refer to Section 7.1.5.1

### **Model Results Presentation**

- Summary table by visit and treatment group (domain scores and total in one output)
- Summary table of change from baseline by treatment group (domain scores and total in one output)
- Listing of LCQ scores by timepoint (baseline and Day 7) and period
- Plot of absolute mean LCQ ±- 95% CI by timepoint and treatment group (4 graphics one for each domain and total score, page by endpoint)
- Summary table of statistical analysis of change from baseline to Day 7 (pre-dose): adjusted posterior medians and 95% credible intervals by treatment, estimated posterior median treatment effect and 90% credible interval, posterior probabilities of interest (difference >0, >1 and >1.3 points on LCQ scale) (page by LCQ endpoint). A difference of 1.3 points is considered to be a minimally important difference.
- Figure of statistical analysis adjusted medians and 95% credible intervals by treatment group (page by LCQ endpoint)

#### **Subgroup Analyses**

Refer to Section 7.1.5.1

#### **Sensitivity and Supportive Analyses**

Refer to Section 7.1.5.1

### 8. SAFETY ANALYSES

The safety analyses will be based on the All Subjects population, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 11: List of Data Displays.

# 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 11: List of Data Displays.

## 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 11: List of Data Displays.

The CSSRS questionnaire will be summarised by the use of a listing, to present data by participant, treatment group and timepoint.

Weight measured during the study will be summarised with standard vitals signs data.

A listing of audiometry changes from baseline will be produced.

#### 9. PHARMACOKINETIC ANALYSES

## 9.1. Primary Pharmacokinetic Analyses

#### 9.1.1. Endpoint / Variables

#### 9.1.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 12.4.3 Reporting Standards for Pharmacokinetic Data).

#### 9.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|------------|--------------------------------|
| Cmax | GSK2798745 for Day 1 and Day 7 |
| Tmax | GSK2798745 for Day 1 and Day 7 |
| AUC(0-3.5) | GSK2798745 for Day 1 and Day 7 |
| C24 | GSK2798745 for Day 8 |

**NOTES:** Additional parameters may be included as required.

### 9.1.2. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

#### 9.1.3. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 9.2. Secondary Pharmacokinetic Analyses

#### 9.2.1. Endpoint / Variables

#### 9.2.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 12.4.3 Reporting Standards for Pharmacokinetic Data).

For atorvastatin, it is expected that patients are on a stable daily dose. Dosing date and time of atorvastatin for Day -1, Day 1, Day 6 and Day 7 will be recorded separately for applicable participants. Therefore, the PKCNC dataset created for atorvastatin will require some non-standard programming to ensure the last dose prior to PK sampling on Day 1 and Day 7 is selected to derive actual sampling times. Time from last dose will therefore vary across participants dependent on when their last dose of atorvastatin was taken.

#### 9.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| Cmax | M1 metabolite for GSK2798745 Day 1 and Day 7 |
| | Atorvastatin and metabolite in available participants Day 1 and Day 7 |
| Tmax | M1 metabolite for GSK2798745 Day 1 and Day 7 |
| | Atorvastatin and metabolite in available participants Day 1 and Day 7 |
| AUC(0-3.5) | M1 metabolite for GSK2798745 Day 1 and Day 7 |
| | Atorvastatin and metabolite in available participants Day 1 and Day 7 |
| C24 | M1 metabolite for Day 8 |
| | Atorvastatin and metabolite in available participants for Day 8 |

**NOTES:** Additional parameters may be included as required.

### 9.2.2. Population of Interest

The secondary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

### 9.2.3. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 10. POPULATION PHARMACOKINETIC (POPPK) AND PHARMACODYNAMIC ANALYSES

Given the sparse plasma sampling scheme for GSK2798745, a non-linear mixed effects methodology will be applied to characterise the population PK of GSK2798745 allowing for the relatively few number of participants. This poppk model will be adapted from a previous model characterised for GSK2798745 in healthy participants [report in progress] to derive some key PK parameter estimates including Cmax, AUC and average concentration of drug over dosing interval (Cav). The influence of participant demographics, baseline characteristics, including baseline disease activity (cough counts), and co-medication on the pharmacokinetics of GSK2798745 in this population will be investigated. The individual participant PK parameters will be estimated and documented for the purposes of any subsequent exposure-response (PK/PD) analyses.

A population systemic exposure-efficacy model will be developed if data permit. Individual PK metrics such as trough concentration observed on Day 8 as well as the estimated average concentration over the dosing interval (Cav) will be used to derive a parametric model quantifying relationship between drug levels and the primary efficacy endpoint (total day-time cough count (10 hours)).

## 10.1. Statistical Analyses / Methods

A summary of the planned population pharmacokinetic analyses are outlined below:

- Drug plasma concentration-time data will be subjected to nonlinear mixed effects modelling using the program NONMEM to develop a population PK model or apply a previous pop pk model developed in healthy participants receiving GSK2798745.
- o Individual post-hoc estimated PK parameters will be summarised descriptively.
- o To support this analysis PopPK and population PK-PD datasets will be generated.

The timeline for these analyses will be independent of statistical analysis complete (SAC). Further details will be documented in a separate CPMS RAP.

The details for the dataset specifications are provided in Appendix 8: Population Pharmacokinetic (PopPK) Analyses.

Detailed Population PK-PD methodology and dataset specifications are presented in Appendix 9: Pharmacokinetic / Pharmacodynamic Analyses.

## 11. REFERENCES

GlaxoSmithKline Document Number.: 2017N31986\_00, A study to assess the effectiveness and side effects of GSK2798745 in participants with chronic cough; 31-MAY-2017.

GlaxoSmithKline Document Number.: 2017N31986\_01, A study to assess the effectiveness and side effects of GSK2798745 in participants with chronic cough; 09-OCT-2017.

GlaxoSmithKline Document Number. : 2017N31986\_02, A study to assess the effectiveness and side effects of GSK2798745 in participants with chronic cough; 22-NOV-2017.

GlaxoSmithKline Document Number.: 2017N31986\_03, A study to assess the effectiveness and side effects of GSK2798745 in participants with chronic cough; 25-JUN-2018.

# 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

A Per Protocol Population is not defined for the study. Important protocol deviations will be summarised and listed.

# 12.2. Appendix 2: Schedule of Activities

## 12.2.1. Protocol Defined Schedule of Events

# **Screening and Follow-up Schedule of Activities**

| Procedure | Screening <sup>1</sup><br>(up to 28 days before<br>Treatment Period 1, Day -1) | Follow up/Early Withdrawal<br>(7-10 days post last dose) | Notes |
|---|---|---|---|
| Informed consent | X | | |
| Inclusion and exclusion criteria | X | | |
| Demography | X | | |
| Medical history (includes substance usage [and family history of premature CV disease]) | Х | | Substances: Drugs, Alcohol, tobacco |
| Full physical exam, including height and weight | X | Х | Height to be measured at screening only. |
| Chest imaging [CXR] | Х | | Not required if chest imaging has been conducted within 12 months of screening with no significant findings. |
| Columbia Suicidality Severity Rating Scale (CSSRS) | Х | Х | Use 'Baseline' CSSRS at Screening. Use the 'Since Last Visit' CSSRS at Follow-up. |
| Human immunodeficiency virus (HIV), hepatitis B (Hep B) and Hepatitis C (Hep C) screen | Х | | |
| Clinical chemistry, haematology and urinalysis (including cardiac troponin) | Х | Х | Non Fasting |
| Follicle-stimulating hormone and estradiol | Х | | As needed in women of non-childbearing potential only. |
| Faecal Occult Blood Test (FOBT) | Х | | FOBT cards will be provided at screening and must be returned to the laboratory and analysed before Day -1. |
| Vital signs (blood pressure, heart rate and temperature) | Х | Х | Triplicate vital signs required at screening. |
| 12-lead ECG | Х | Х | Triplicate ECG required at screening. |
| Forced Expiratory Volume in One Second (FEV1) | Х | | Not required if documented evidence of FEV1 ≥ 80% within the 6 months before screening. |
| Procedure | Screening <sup>1</sup> | Follow up/Early Withdrawal | Notes |
|---|---|---|---|
| | (up to 28 days before<br>Treatment Period 1, Day -1) | (7-10 days post last dose) | |
| Cough Severity & Urge to Cough Visual Analogue Scale (VAS) | X (Severity only) | X (Severity & Urgency) | Urge to cough VAS will not be completed at screening. |
| Audiometry | | X | Audiometry to be done anytime between end of Treatment Period 2 and Follow-up. |
| Concomitant Medication review | X | Х | |
| Adverse event (AE)/serious adverse event (SAE) review | Х | X | SAEs collected from the time of consent. AEs collected from the time of first dose. |

<sup>1.</sup> Screening assessments may be conducted at multiple visits, if required, but all samples for laboratory safety tests to be collected at one visit (unless repeats).

### **Treatment Period 1 and 2 Schedule of Activities**

| Procedure | Treatment Period 1 and 2 (Washout 14-21 days) | | | | | Notes |
|---|---|---|---|---|---|---|
| Procedure | Day -1 | Day 1 | Day 2-6 | Day 7 | Day 8 | Notes |
| Study Treatment | | | | | | |
| Randomisation | | X (TP1 only) | | | | Can be done on Day –1 or Pre-dose Day 1. Participants will be stratified based on inclusion in a cough study within the last 12 months (defined as taking an investigational product in a cough study within the last 12 months). |
| Study Treatment dispensed | | Х | | | | |
| Study Treatment dosing | | Х | X | Х | | Home dosing on Days 2-6. Dosing to be at about the same time each day ( $\pm$ 2 hours relative to dosing on Day 1). |
| Diary Card dispensed | | Х | | X (TP1 only) | | Diary card used to collect dosing information, AEs and concomitant medications. Diary card dispensed on Day 7 in Treatment Period 1 only (to collect AEs and concomitant medications during washout period). |

| Day and day | T | reatment Period | d 1 and 2 (Was | N. C. | | |
|---|---|---|---|---|---|---|
| Procedure | Day -1 | Day 1 | Day 2-6 | Day 7 | Day 8 | - Notes |
| Efficacy Assessments | | | | | | |
| 24- hour Cough Counting Starts | Х | | | X | | On Day 7, the cough counter must be attached immediately after dosing. Participant to be advised to avoid noisy environments whilst wearing the counter, and to stay awake for 10 h after attachment of cough monitor. |
| 24- hour Cough Counting Ends | | X | | | Х | On Day 1, the cough counter must be removed before dosing. |
| Cough Severity & Urge to Cough VAS | Х | | | X (pre-dose) | | To be completed before other assessments |
| Leicester Cough Questionnaire (LCQ) | Χ | | | X (pre-dose) | | To be completed before other assessments |
| Safety Assessments | | | | | | |
| Brief physical exam | Χ | | | | Х | Baseline can be done on Day –1 or Pre-dose Day 1 |
| Weight | Χ | | | | Х | Baseline can be done on Day –1 or Pre-dose Day 1 |
| Vital signs (blood pressure, heart rate and temperature) | | X (pre-dose) | | | Х | Single measurements |
| 12-lead ECG | | X (pre-dose) | | | Х | Single measurements |
| Clinical chemistry, haematology and urinalysis (including cardiac troponin) | | X (pre-dose) | | | Х | Non-fasting. |
| FOBT | | | | Х | | FOBT cards will be provided on Day 1 and returned on Day 7 or 8, if possible (or returned by post). |
| CSSRS | X | | | | Х | Use the 'Since Last Visit' CSSRS questionnaire. The pre-dose CSSRS in each Treatment Period can be done on Day –1 or Pre-dose Day 1. |

| Dreadure | T | reatment Perio | d 1 and 2 (Was | ys) | Notes | |
|---|---|---|---|---|---|---|
| Procedure | Day -1 | Day 1 | Day 2-6 | Day 7 | Day 8 | Notes |
| Audiometry | X | | | | | Pre-Treatment Period 1 audiometry can be done anytime between Screening and Treatment Period 1, Day 1, pre-dose. Pre-Treatment Period 2 audiometry can be done any time during the washout period (up to Treatment Period 2, Day 1 pre-dose). |
| Concomitant Medication review | Х | Х | Х | Х | Х | Concomitant medications collected in Diary Card during washout period. |
| SAE/AE review | X | Х | Х | Х | Х | AEs collected in Diary Card during washout period. |
| Other Assessments | | | | | | |
| PK blood samples | | Х | | Х | Х | Day 1 and Day 7: predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5 h post dose Day 8: 24 h post dose For participants taking atorvastatin, an extra sample will be taken at each time-point. |
| Optional Genetic Sample | | Х | | | | Can be taken any time after consent has been signed and the participant has been randomised. |

- The Cough Severity & Urge to Cough VAS should be completed before the LCQ, and both questionnaires should be completed before any other assessments.
- When scheduled at the same time-points, 12-lead ECGs and vital signs should be completed before any blood draws.
- The timing of assessments should allow PK samples to be taken as close as possible to the nominal time-point.
- The timing and number of planned study assessments, including: safety and pharmacokinetic assessments may be altered during the course of the study based on newly available data (e.g. to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.
- Any changes in the timing or addition of time points for any planned study assessments must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The IRB/IEC will be informed of any safety issues that require alteration of the safety monitoring scheme or amendment of the ICF.

# 12.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

### 12.3.1. Study Phases and Treatment Emergent Rules for AEs

This study is a multiple dose two period crossover study. As such, AEs will be attributed to the treatment received within the relevant study period based on the dates of the AEs in relation to dosing date. This is as per IDSL dataset standards. This is detailed in the table below.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date (Period 1) |
| On-Treatment (Period 1) | If AE Start Date is on or after Study Treatment Start Date (Period 1) & before Study Treatment Start Date (Period 2). |
| | Study Treatment Start Date (Period 1) ≤ AE Start Date < Study Treatment Start Date (Period 2) |
| On-Treatment (Period 2) | If AE Start Date is on or after Study Treatment Start Date (Period 2) & before Follow-<br>Up. |
| | Study Treatment Start Date (Period 2) ≤ AE Start Date ≤ Follow-Up Date |
| Post-Treatment | If AE Start Date is on or after Follow-Up. |
| | AE Start Date > Follow-Up Date |

#### NOTES:

• Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

### 12.3.1.1. Study Phases for Concomitant Medication

This study is a multiple dose two period crossover study. As such, Concomitant Medications will be attributed to the treatment received within the relevant study period based on the dates of the AEs in relation to dosing date. This is as per IDSL dataset standards. This is detailed in the table below.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | CM Start Date < Study Treatment Start Date (Period 1) |
| On-Treatment<br>(Period 1) | If CM Start Date is on or after Study Treatment Start Date (Period 1) & before Study Treatment Start Date (Period 2). Study Treatment Start Date (Period 1) ≤ CM Start Date < Study Treatment Start Date (Period 2) |
| On-Treatment<br>(Period 2) | If CM Start Date is on or after Study Treatment Start Date (Period 2) & before Follow-Up. Study Treatment Start Date (Period 2) ≤ CM Start Date ≤ Follow-Up Date |

# 12.4. Appendix 4: Data Display Standards & Handling Conventions

### 12.4.1. Reporting Process

| Software | Software |
|---|---|
| The currently sup- | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : UK1SALX00175.corpnet2.com |
| HARP Compound | : \ARPROD\GSK2798745\207702\Internal_01 |
| | : \ARPROD\ GSK2798745\207702\Final_01 |
| <b>Analysis Datasets</b> | Analysis Datasets |
| <ul> <li>Analysis datasets will be created according to Legacy GSK A&amp;R dataset standards (Integrated Data<br/>Standards Library).</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for the Final reporting effort. | |

### 12.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

Unscheduled visits will not be included in summary tables and/or figures.

| All unscheduled v | All unscheduled visits will be included in listings. |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | ontinuous Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | gorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

# 12.4.3. Reporting Standards for Pharmacokinetic Data

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to GUI_51487. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Pop-PK file (CSV format) for the POP-PK analysis by CPMS will be created by S&P according to the data specification detailed in Section 12.8.2 Population Pharmacokinetic (PopPK) Dataset Specification. |
| NONMEM/PK/PD<br>File | PK/PD file (CSV format) for the PK/PD analysis by CPMS will be created by S&P according to the data specification detailed in Section 12.9.2 Pharmacokinetic/Pharmacodynamic Dataset Specification. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameters to be Derived | The following PK parameters will be derived by CPMS: Non Compartmental (to be forwarded to Statistics and Programming): Cmax, Tmax and AUC(0-3.5), C24 on Day 8 PopPK parameters include CL/F, AUC(0-24), Cav and Cmax |
| Pharmacokinetic Para | Pharmacokinetic Parameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters, December 2009. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |

### 12.5. Appendix 5: Derived and Transformed Data

#### 12.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

### 12.5.2. Study Population

#### **Treatment Compliance**

• In this study, participants take 2 tablets on Day 1 (2 x 2.4 mg) and 1 tablet (1 x 2.4 mg) on Days 2 through to 7, therefore treatment compliance will be calculated based on the formula:

Treatment Compliance = Number of Actual Doses / Planned Number of Doses,

which will be calculated as,

#### [No. of tablets taken / (No. of days in period + 1)] \* 100,

where No. of days in period = (Date of last dose- Date of first Dose) +1 in each period. The denominator has 1 added to it to account for the fact that 2 tablets are taken on Day 1 and 1 tablet is taken on all other days.

- Treatment compliance could be greater than 100% if there are events of overdose as recorded for 'tablets taken'.
- Reasons for treatment not being returned will be recorded (tick box on eCRF).
- Compliance during each study period will be calculated.
- For each study period, a bottle containing 15 tablets is dispensed. At the end of each period, 7 tablets should remain if a participant has taken all medication correctly and returned unused tablets correctly.

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

Cumulative Dose = Sum of (Number of Days on 4.2 mg x Total Daily Dose (for 4.2 mg)) + Sum of (Number of Days on 2.4 mg x Total Daily Dose (for 2.4 mg))

### **Treatment Compliance**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

### 12.5.3. **Efficacy**

### Total Cough Counts at 10h and 24h

- Variance stabilising transformations (e.g. taking natural logarithms of the observed responses) may be implemented, if deemed necessary by the study statistician. If transformations are used the results will be reported on the back-transformed response scales.
- Other efficacy endpoints to be statistically analysed will also be assessed for data transformation

### 12.5.3.1. Cough Count SI and A&R Dataset Specifications

### **SI Dataset COUGH**

Provided by Data Management, this is based on data provided by Vitalograph in file 207702 cough YYYYMMDD.csv

| Column<br>Name | Data<br>Type/Format | Label (additional detail from transfer agreement) |
|---|---|---|
| STUDYID | Char 10 | Unique identifier for the study |
| SUBJID | Num 10. | Subject ID |
| VISIT | Char 40 | Visit description |
| VISITNUM | Num 7.2 | Visit sequence number |
| PTM | Char 40 | Planned timepoint description |
| PTMNUM | Num 7.2 | Planned timepoint sequence number |
| CENTREID | \$45 | Centre ID |
| ACTDT | Date9. | Actual date of assessment (Start date of cough monitoring) |
| ACTSTTM | Time8. | Actual start time of assessment (Start time of the Cough Monitoring in 24 hour format) |
| ENTM | Time5. | Stop time (Stop time of the Cough Monitoring in 24 hour format) |
| COVEID | \$80 | Cough vendor ID |
| COVEIDC | \$8 | Cough vendor ID code |
| EVNTDT | Date9. | Event date (Event date in DDMMMYYYY format) |
| EVNTTM | Time5. | Event time (Event time in 24 hour format displayed as HH:MM. This is the time with the seconds and milliseconds removed) |
| PRREFID | Char 20 | Procedures reference ID (Sample ID (unique ID) – The serial number from CF Card) |
| ELTIMES | Num 8.3 | Elapsed time, in seconds (The seconds and milliseconds portion of the event time displayed as SS.MMM. This combined with EVTDT and EVNTTM will provide the full date and time of the cough event) |

### External Dataset g207702 session YYYYMMDD.sas7bdat

Provided by Vitalograph directly to Statistics and Programming. To be merged with SI COUGH dataset to derive missing data periods.

| Column<br>Name | Data Type /<br>Format | Description / Notes |
|---|---|---|
| STUDYID | CHAR 6 | Study Protocol ID – 207702 |
| SUBJID | CHAR 6 | The 6 digit Subject ID. |
| VISIT | CHAR 23 | The name of the visit. |
| VISITNUM | CHAR 7 | Visit sequence number. |
| CENTREID | CHAR 6 | The 6 digit Site ID. |
| ACTDT | CHAR 9 | Start date of the Cough Monitoring in the format DDMMMYYYY. |
| ACTSTTM | CHAR 5 | Start time of the Cough Monitoring in 24 hour format displayed as HH:MM. |
| ENTM | CHAR 5 | Stop time of the Cough Monitoring in 24 hour format displayed as HH:MM. |
| COVEID | CHAR 80 | To be populated with 'Vitalograph Business Park, Maids Moreton, BUCKINGHAM, MK18 1SW' |
| COVEIDCD | CHAR 8 | To be populated with 0001 |
| PRREFID | CHAR 6 | The Card Serial Number |
| FIELD_NAME | CHAR 100 | "Session Status" for the status of the session row, each session will display this row e.g. Accepted. |
| NOEVNEDT | CHAP 20 | The following event rows will only appear for sessions that have these events recorded. The label associated to the non-cough event will be displayed using: "Sleep" — Sleep start event type "Wake" — Wake event type, will be set to the end of the recording if the subject did not wake during the session "Removal" — Removed device event type "Restore" — Restored device event type, will be set to the end of the recording if the device is never restored "Early termination" — The session is terminated early, possibly due to a CF card or battery failure. "Early Stoppage" — The session is stopped when the clinic or subject stops the device manually. "Late Attachment" — The device is attached late. "Flagged Area Start" — Flagged area start event type "Flagged Area End" — Flagged area end event type See cough analysis plan (Vitalograph) for further details. |
| NCEVNTDT | CHAR 30 | Date of the non-cough event. For sessions that have been rejected, 'Rejected' will be displayed. For sessions that have been accepted with no events, 'Accepted with no events' will be displayed. For sessions that have been accepted with events, the full date and time of the event will be displayed including milliseconds, e.g. 10JUL2017 01:17:00:410. |

### **A&R dataset COUGHALL**

This derived dataset will include the original SI COUGH data merged together with the session data (transposed event dates/times) to provide all event dates/times in a format suitable for calculation of time periods. This dataset will not need to be formally QCd, but will be available as an intermediate dataset. QC of the dataset COUGHTOT will provide a QC that the non cough-events have merged and been used correctly.

| Column<br>Name | Data Type /<br>Format | Label (additional detail from data transfer agreement) |
|---|---|---|
| STUDYID | Char 10 | Unique identifier for the study |
| SUBJID | Num 10. | Subject ID |
| VISIT | Char 40 | Visit description |
| VISITNUM | Num 7.2 | Visit sequence number |
| PTM | Char 40 | Planned timepoint description |
| PTMNUM | Num 7.2 | Planned timepoint sequence number |
| CENTREID | \$45 | Centre ID |
| ACTDT | Date9. | Actual date of assessment |
| | | (Start date of cough monitoring) |
| ACTSTTM | Time8. | Actual start time of assessment |
| | | (Start time of the Cough Monitoring in 24 hour format) |
| ENTM | Time5. | Stop time |
| | | (Stop time of the Cough Monitoring in 24 hour format) |
| COVEID | \$80 | Cough vendor ID |
| COVEIDCD | \$8 | Cough vendor ID code |
| EVNTDT | Date9. | Event date |
| | | (Event date in DDMMMYYYY format) |
| EVNTTM | Time5. | Event time |
| | | (Event time in 24 hour format displayed as HH:MM. This |
| | | is the time with the seconds and milliseconds removed) |
| PRREFID | Char 20 | Procedures reference ID |
| | | (Sample ID (unique ID) – The serial number from CF |
| EL TIMEO | NI OO | Card) |
| ELTIMES | Num 8.3 | Elapsed time, in seconds |
| | | (The seconds and milliseconds portion of the event time |
| | | displayed as SS.MMM. This combined with EVTDT and |
| | | EVNTTM will provide the full date and time of the cough |
| STOPDT | Date9. | event) |
| 310001 | Dates. | Event stop date (DERIVED VARIABLE – merge on last cough event and |
| | | select date of event, should be the next calendar day if |
| | | 24 hour monitoring achieved) |
| EVNDTTM | Datetime20. | Cough event date and time |
| LVINDITIVI | Datelinezo. | (DERIVED VARIABLE – merge together each cough |
| | | date, time and seconds and apply format) |
| STADTTM | Datetime20. | Cough monitoring start date and time |
| 317.511111 | 3 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 | (DERIVED VARIABLE – merge together start date, time |
| | | and seconds and apply format) |
| STODTTM | Datetime20. | Cough monitoring stop date and time |
| | | ( <b>DERIVED VARIABLE</b> – merge together stop date, time |
| | | and seconds and apply format) |
| | L | 117 -7 |

| Column | Data Type / | Label (additional detail from data transfer agreement) |
|---|---|---|
| Name | Format | Florand area start data and time |
| FAREAS | Datetime20. | Flagged area start date and time |
| | | (DERIVED VARIABLE – convert character date variable |
| EADEAE | D 1 1 1 2 2 2 2 2 | provided to numeric date format) |
| FAREAE | Datetime20. | Flagged area stop date and time |
| | | ( <b>DERIVED VARIABLE</b> – convert character date variable provided to numeric date format) |
| ASLEEP | Datetime20. | Sleep period start date and time |
| ASLEEP | Datetimezo. | ( <b>DERIVED VARIABLE</b> – convert character date variable |
| | | provided to numeric date format) |
| AWAKE | Datetime20. | Sleep period stop date and time |
| AVVAIL | Datetimezo. | ( <b>DERIVED VARIABLE</b> – convert character date variable |
| | | provided to numeric date format) |
| EARLYTRM | Datetime20. | Early termination date and time |
| LAIXLIIIXW | Datelinezo. | ( <b>DERIVED VARIABLE</b> – convert character date variable |
| | | provided to numeric date format) |
| REMOVE | Datetime20. | Removal date and time |
| INLINIOVE | Datelinezo. | ( <b>DERIVED VARIABLE</b> – convert character date variable |
| | | provided to numeric date format) |
| RESTOR | Datetime20. | Restore date and time |
| | | ( <b>DERIVED VARIABLE</b> – convert character date variable |
| | | provided to numeric date format) |
| EARLYSTO | Datetime20. | Early stoppage date and time |
| | | ( <b>DERIVED VARIABLE</b> – convert character date variable |
| | | provided to numeric date format) |
| LATEATT | Datetime20. | Late attachment date and time |
| | | ( <b>DERIVED VARIABLE</b> – convert character date variable |
| | | provided to numeric date format) |
| STATUS | Char 120. | Status of cough recording |
| TRTCD | Num 8 | Randomised Treatment Code (Seq) |
| TRTGRP | Char 120. | Randomised Treatment Group (Seq) |
| ATRTCD | Num 8 | Actual Treatment Code (Seq) |
| ATRTGRP | Char 120. | Actual Treatment Group (Seq) |
| PTRTCD | Num 8 | Period Treatment Code |
| PTRTGRP | Char 120. | Period Treatment Group |
| PATRTCD | Num 8 | Period Actual Treatment Code |
| PATRTGRP | Char 120. | Period Actual Treatment Group |

Note: If there is more than one sleep period, then name subsequent sleep and awake events as ASLEEP1, ASLEEP2, AWAKE1, AWAKE2 etc. The same logic would apply to more than one removal/restore or flagged area.

### **A&R dataset COUGHTOT**

This dataset will use A&R dataset COUGHALL and create hourly, 10h and 24h counts with missing data periods imputed where appropriate. Log transformed variables to be included for use in the analysis.

| Column<br>Name | Data Type /<br>Format | Label (additional detail from data transfer agreement) |
|---|---|---|
| STUDYID | Char 10 | Unique identifier for the study |

| Column | Data Type / | Label (additional detail from data transfer |
|---|---|---|
| Name | Format | agreement) |
| SUBJID | Num 10. | Subject ID |
| VISIT | Char 40 | Visit description |
| VISITNUM | Num 7.2 | Visit sequence number |
| PTM | Char 40 | Planned timepoint description |
| PTMNUM | Num 7.2 | Planned timepoint sequence number |
| CENTREID | \$45 | Centre ID |
| Hourly, 10h and | Datetime20. | |
| FLAGHR | Datetime20. | Timepoint Flag (DERIVED VARIABLE – one row per hourly interval, 10h, overall 24 period, plus one row for each of the 3 intervals within the 24h period) Values are: 1 2 |
| | | 23 24 100 /*for 10h*/ 240 /*for 24h*/ 499 /*for awake period 1*/ 500 /*for sleep period*/ 501 /*for awake period 2*/) 1120 /*for first 12h*/ 1080 /*for next 8h*/ 1040 /*for next 4h*/ |
| FLAGHRC | Char 10 | Timepoint Flag Description (DERIVED VARIABLE – as above, one row per hourly interval, 10h, overall 24 period, plus one row for each of the 3 intervals within the 24h period) Character values are: 0-1h 1-2h 22-23h 23-24h 10h 24h 24h Awake1 24h Awake1 24h Sleep1 24h Awake2 24h 0-12h 24h 12-20h 24h 20-24h |
| Imputation der | ivation variable | - |
| FLAGIMP | Char 2 | Flag Imputed (DERIVED VARIABLE) Values are: Y /*Yes imputed value*/ YR /*Yes imputed but based on full 24h as an individual interval does not meet 60% criteria, but full 24h does */ |

| Column | Data Type / | Label (additional detail from data transfer |
|---|---|---|
| Name | Format | agreement) |
| | | NA /*Not applicable – cannot be imputed due to 60% |
| | | rule */ |
| | | ' ' data complete and not imputed |
| Stratification v | <u>rariables</u> | |
| PRIOR | Char 1 | Prior cough study participation |
| | | (Renamed SCHORSCD variable in SC dataset) |
| | | Y=Yes, N=No for answer to stratification question |
| PRIORCD | Num 8 | Numeric code for prior study participation |
| | | (Derived, if PRIOR=Y then PRIORCD=1 else if |
| D-4-14: | | PRIOR=N then PRIORCD=2) |
| | nt variables from | |
| STADTTM | Datetime20. | Cough monitoring start date and time (from COUGHALL) |
| STODTTM | Datetime20. | Cough monitoring stop date and time |
| | | (from COUGHALL) |
| FAREAS | Datetime20. | Flagged area start date and time |
| | Detetimen | (from COUGHALL) |
| FAREAE | Datetime20. | Flagged area stop date and time (from COUGHALL) |
| ASLEEP | Datetime20. | Sleep period start date and time |
| ASLEEF | Datetimezo. | (from COUGHALL) |
| AWAKE | Datetime20. | Sleep period stop date and time |
| / (V / (I (L | Batetime20. | (from COUGHALL) |
| EARLYTRM | Datetime20. | Early termination date and time |
| | | (from COUGHALL) |
| REMOVE | Datetime20. | Removal date and time |
| | | (from COUGHALL) |
| RESTOR | Datetime20. | Restore date and time |
| | | (from COUGHALL) |
| EARLYSTO | Datetime20. | Early stoppage date and time |
| | | (from COUGHALL) |
| LATEATT | Datetime20. | Late attachment date and time |
| 0 | -4-1 | (from COUGHALL) |
| COLICHTOT | | Cough Count Total Day |
| COUGHTOT | Num 8 | Cough Count Total Raw (DERIVED VARIABLE – create for each hourly interval |
| | | and for 10h and 24h period) |
| COUGHIMP | Num 8 | Cough Count Total Imputed |
| COOCI IIIVII | Numo | (DERIVED VARIABLE – create for each hourly interval |
| | | and for 10h and 24h period, imputation based on rules |
| | | as per RAP) |
| Log transform | ed cough coun | t total variables |
| LOGCTOT | Num 8 | Log transformed cough total |
| LOGCIMP | Num 8 | Log transformed imputed cough total |
| Subject baseli | ne derivation v | <u>ariables</u> |
| CTOTBS | Num 8 | Subject baseline |
| CIMPBS | Num 8 | Imputed subject baseline |
| CTOTBP1 | Num 8 | Baseline period 1 |
| CTOTBP2 | Num 8 | Baseline period 2 |

| Column<br>Name | Data Type /<br>Format | Label (additional detail from data transfer |
|---|---|---|
| CIMPBP1 | Num 8 | agreement) Imputed baseline period 1 |
| CIMPBP2 | Num 8 | Imputed baseline period 2 |
| | | vation variables |
| CTOTPA | Num 8 | Period adjusted baseline |
| CIMPPA | Num 8 | Period adjusted imputed baseline |
| Log transforme | ed subject base | eline derivation variables |
| LCTOTBS | Num 8 | Log transformed subject baseline |
| LCIMPBS | Num 8 | Log transformed imputed subject baseline |
| Log transformed period adjusted baseline derivation variables | | |
| LCTOTPA | Num 8 | Log transformed period adjusted baseline |
| LCIMPPA | Num 8 | Log transformed period adjusted imputed baseline |
| Standard treate | ment group var | riables |
| TRTCD | Num 8 | Randomised Treatment Code (Seq) |
| TRTGRP | Char 120. | Randomised Treatment Group (Seq) |
| ATRTCD | Num 8 | Actual Treatment Code (Seq) |
| ATRTGRP | Char 120. | Actual Treatment Group (Seq) |
| PTRTCD | Num 8 | Period Treatment Code |
| PTRTGRP | Char 120. | Period Treatment Group |
| PATRTCD | Num 8 | Period Actual Treatment Code |
| PATRTGRP | Char 120. | Period Actual Treatment Group |

### 12.5.3.2. Cough Count Missing Data Period Algorithms

### **Codes:**

L = Low hour, H=High hour, M=missing time period

X = Start of missing period (e.g. removal), Y = End of missing period (e.g. restore)

LA = Late attachment ET = Early Termination ES = Early Stoppage

S = Beginning of sleep period

A = End of sleep period (awakening)

All measured in seconds e.g. 1h = 3600 seconds

X, Y, S, A, LA, ET and ES represent time from start of cough monitoring in seconds Shaded areas represent potential missing data time intervals

A1 =first awake interval, S1 =sleep interval, A2 =second awake interval

### 1. HOURLY COUGH COUNT TOTALS

a. Missing periods with a start and end (removal/restore, flagged start/flagged stop)



If  $X \le L$  then do; If  $Y \le H$  then M = Y - L

Else if Y > H then M = H - L (should be 3600 secs)

If  $L \le X \le H$  then do; If  $Y \le H$  then M = Y - X

Else if Y > H then M = H - X

b. Late attachment, early termination or early stoppage

 Oh
 1h
 2h

 (L)
 (H)

 LA
 ET/ES

 LA
 ET/ES

If 
$$L \le LA \le H$$
 then  $M = (H - L) - (H - LA)$ ,  
Else if  $LA > H$  then  $M=H-L$ 

If 
$$L \le ET \le H$$
 then  $M = H - ET$  (same for ES),  
Else if  $ET \le L$  then  $M=H-L$ 

### 2. 10H DAYTIME COUGH COUNT TOTALS

a. Missing periods with a start and end (removal/restore, flagged start/flagged stop, sleep/awake)





If 
$$X < 36000$$
 then do; If  $Y <= 36000$  then  $M = Y - X$   
Else if  $Y > H$  then  $M = 36000 - X$ 

If LA 
$$<$$
 36000 then M = LA  
If ET  $<$  36000 then M = 36000 – ET (same for ES)

### 3. 24H COUGH COUNT TOTALS

a. Awake Period 1 (A1) {or first 12h (0-12h) if applicable}



If 
$$X \le S$$
 then do; If  $Y \le S$  then  $M = Y - X$   
Else if  $Y \ge S$  then  $M = S - X$ 



If 
$$LA < S$$
 then  $M = LA$   
If  $ET/ES < S$  then  $M = S - ET/ES$ 

b. Sleep Period (S1) {or next 8h (12-20h) if applicable}

 Oh
 A1
 S
 S1
 A
 A2
 24h

 X
 Y
 Y</

If X < S then do; If  $S \le Y \le A$  then M = Y - S

Else if Y > A then M = A - S (sleep period)

If  $S \le X \le A$  then do; If  $Y \le A$  then M = Y - X

Else if Y > A then M = A - X

0h A1 S S1 A A2 24h

LA | ET |

If  $S \le LA \le A$  then M = LA - SIf  $S \le ET/ES \le A$  then M = A - ET/ES

c. Awake Period 2 (A2) {or last 4h (20-24h) if applicable}

0h A1 S S1 A A2 24h X Y X Y

If X < A and Y > A then M = Y - AElse if X >= A then M = Y - X

0h A1 S S1 A A2 24h

LA ET

If  $A \le LA \le 24h$  then M = LA - AIf  $A \le ET/ES \le 24h$  then M = 86460 - ET/ES

Note: Value in seconds for 24 hours has 60 seconds added to allow for discrepancies between date/time variables that do/do not include seconds.

#### 12.5.3.3. Cough Count Imputation Derivations

Imputation of cough counts will be applied when at least 60% of the cough monitoring time is present. If less than 60% of data is available then the missing time period will not be imputed (with the exception of the overall 24h scenario described in Section 7.2.2). Imputed cough counts within each time period of interest (hourly, 10h, 24h) will be calculated as follows:

$$imputed\ cough\ count\ (COUGHIMP) \\ = integer\ \Big[ cough\ count\ (COUGHTOT) \\ + \left( missing\ proportion\ * \Big\{ \frac{cough\ count\ (COUGHTOT)}{1-missing\ proportion} \Big\} \Big) \Big]$$

For example during the 10h period, if we have 3 hours of missing cough monitoring and the databased cough count for the remaining 7 hours is 500 then the imputed cough count would be:

imputed cough count = integer 
$$\left[500 + \left(0.3 * \left\{\frac{500}{1 - 0.3}\right\}\right)\right]$$
  
imputed cough count = integer  $\left[500 + 214.29\right] = 714$ 

#### 12.5.4. Pharmacokinetic

#### **Pharamacokinetic Parameters**

- Observed Cmax
- Observed AUC(0-3.5)
- Observed C24 Day 8
- Observed Tmax

### 12.5.5. Population Pharmacokinetic (PopPK)

#### **Estimated PK Parameters from PopPK Analyses**

- Model-based Cav (Average conc over 24h)
- Model-based AUC(0-24)
- Model-based Cmax
- Model-based CL/F

Note: produced as part of the PopPK analyses and independent of SAC

# 12.5.6. Operating Characteristics of Decision Criteria Based on Conditional Probabilities

Operating characteristics for the decision criteria were produced based on 10000 simulations to show the long-run properties of the decision rules for a variety of assumptions. For the positive criterion the operating characteristics answer the question "if we ran the study 10000 times, what percentage of those studies would declare a

positive result for the specified set of assumptions?". For the negative criterion the operating characteristics answer the question "if we ran the study 10000 times, what percentage of those studies would declare a negative result for the specified set of assumptions?".

#### **Positive Criterion**

The figure below shows operating characteristics for a range of true treatment ratios and final sample sizes, using the variability assumed for the protocol (0.280). This figure shows the percentage of studies giving a 90% conditional probability of a positive study at the final analysis, conditioning on a treatment ratio of 0.5 (very good effect) for the post-interim data.

The **blue/circle** line shows the operating charateristics if the true treatment ratio was 0.5. If the assumptions are true, a final sample size of 24 would give **86.04%** of studies having at least 90% conditional probability of declaring a positive result when the variability from the protocol is assumed. If the true treatment ratio is 1 (**purple/diamond** line) only **1.78%** of studies would have at-least 90% conditional probability of declaring a postive result.





Similar plots were produced based on variability 80% and 120% of that assumed for the protocol and showed changes to these results as expected (data not shown). For example, assuming a smaller variance of 0.179 and larger variance of 0.403 and a true treatment ratio of 0.5, a final sample size of 24 would give **97.05%** and **71.45%** of studies,

respectively, having at least 90% conditional probability of declaring a positive result. Assuming a smaller variance of 0.179 and larger variance of 0.403 and a true treatment ratio of 1, a final sample size of 24 would give **1.63%** and **1.82%** of studies, respectively, having at least 90% conditional probability of declaring a positive result.

#### **Negative Criterion**

The figure below shows operating characteristics for a range of true treatment ratios and final sample sizes, using the variability assumed for the protocol (0.280). This figure shows the percentage of studies giving a 90% conditional probability of a negative study at the final analysis, conditioning on a treatment ratio of 0.90 (minimal effect) for the post-interim data.

The **purple/diamond** line shows the operating charateristics if the true treatment ratio was 1.0. If the assumptions are true, a final sample size of 24 would give **78.68%** of studies having at least 90% conditional probability of declaring a negative result when the variability from the protocol is assumed. However, if the true treatment ratio is 0.5 (**blue/circle** line) only **0.57%** of studies would have at-least 90% conditional probability of declaring a negative result.





Similar plots were produced based on variability 80% and 120% of that assumed for the protocol and showed changes to these results as expected (data not shown). For example, assuming a smaller variance of 0.179 and larger variance of 0.403 and a true treatment ratio of 1.0, a final sample size of 24 would give **93.44%** and **62.44%** of studies,

respectively, having at least 90% conditional probability of declaring a negative result. Assuming a smaller variance of 0.179 and larger variance of 0.403 and a true treatment ratio of 0.5, a final sample size of 24 would give **0.45%** and **0.75%** of studies, respectively, having at least 90% conditional probability of declaring a negative result.

### 12.6. Appendix 6: Reporting Standards for Missing Data

### 12.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Participant study completion (i.e. as specified in the protocol) was defined as a participant who has completed all phases of the study, including the follow-up visit. |
| | <ul> <li>Withdrawn participants will not be replaced in the study</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 12.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered<br/>to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| Total cough counts (10h, 24h, hourly) | <ul> <li>Consideration will be given to instances where the monitor is turned off<br/>unexpectedly, or where a participant has a sleep period recorded during the<br/>primary day-time hours 10h period.</li> </ul> |
| | <ul> <li>Vitalograph will provide a session acceptance file that will details removal ar<br/>restore dates/times of the monitor for each session (e.g. period 1 day -1)</li> </ul> |
| | See Section 7.1.1 for further details on pro-rated data imputation. |
| Severity and Urge to Cough (VAS) | Missing data will not be replaced |
| LCQ | Missing data will not be replaced |

## 12.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | Start and End dates for adverse events must be complete in the eCRF. |
| Concomitant<br>Medications/<br>Medical History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

### 12.7. Appendix 7: Values of Potential Clinical Importance

### 12.7.1. Laboratory Values

| Hematology | | | |
|---|---|---|---|
| Analyte | Effect | Relative – Low<br>(Multipliers of LLN) | Relative – High<br>(Multipliers of ULN) |
| White Blood Cell Count (x109/ L) | | 0.67 | 1.82 |
| Neutrophil Count (x10 <sup>9</sup> / L) | | 0.83 | |
| | Male | | 1.03 |
| Hemoglobin (g/L) | Female | | 1.13 |
| Hamatacrit (ratio of 1) | Male | | 1.02 |
| Hematocrit (ratio of 1) | Female | | 1.17 |
| Platelet Count (x109/ L) | | 0.67 | 1.57 |
| Lymphocytes (x10 <sup>9</sup> / L) | | 0.81 | |
| Monocytes (x10 <sup>9</sup> / L) | | 0.5 | 1.8 |
| Red Blood Cell Count (x109/ L) | | 0.7 | 1.7 |
| Reticulocytes (%) | | 0 | 1.5 |

| Chemistry | | | |
|---|---|---|---|
| Analyte | Effect | Relative – Low<br>(Multipliers of LLN) | Relative – High<br>(Multipliers of ULN) |
| Calcium (mmol/L) | | 0.91 | 1.06 |
| Glucose (mmol/L) | | 0.71 | 1.41 |
| Potassium (mmol/L) | | 0.86 | 1.10 |
| Sodium (mmol/L) | | 0.96 | 1.03 |
| Blood Urea Nitrogen (mmol/L) | | 0.7 | 1.5 |
| Total Protein (mg/dL) | | 0.6 | 1.7 |
| Creatinine phosphokinase (IU/L) | | 0 | 1.8 |
| Direct Bilirubin (umol/L) | | 0 | 1.6 |
| Analyte | Effect | Relative – Low<br>(Absolute Value) | Relative – High<br>(Absolute Value) |
| Creatinine (umol/L) | Chg from Baseline | | > 44 umol/L |
| Cardiac Troponin I (ug/L) | | | 0.09 ug/L |
| FOBT | | Positive | Positive |

**Urinalysis:** During the study, a dipstick result (positive or negative) will be recorded for each participant at each relevant timepoint. If the dipstick result is positive, a microscopy will be performed. The urinalysis dipstick result at Day 8 will be compared with Day 1

(Pre Dose) and data of PCI will be flagged where a result changes from negative to positive and/or a microscopy is performed.

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5x ULN |
| | umol/l | | ≥ 1.5x ULN T.Billirubin |
| T. Bilirubin + ALT | μmol/L,<br>U/L | High | + |
| | U/L | | ≥ 2x ULN ALT |

### 12.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | • | | |
| Absolute QTc Interval | msec | | >500 |
| Absolute PR Interval | msec | <110 | >220 |
| Absolute QRS Interval | msec | <75 | >110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >60 |

# 12.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Cor | ncern Range |
|--------------------------|-------|--------------|-------------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >160 |
| Diastolic Blood Pressure | mmHg | <45 | >100 |
| Heart Rate | bpm | <40 | >110 |

| Vital Sign Parameter | Units | | Clinical Con | inical Concern Range | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decr | ease | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

### 12.8. Appendix 8: Population Pharmacokinetic (PopPK) Analyses

### 12.8.1. Population Pharmacokinetic (PopPK) Methodology

#### 12.8.1.1. Software

All analysis will be performed in the validated Modelling and Analysis Platform (MAP). MAP consists of a Linux desktop containing various modelling applications, including NONMEM, PsN, Pirana, R and RStudio. All software versions used will be documented.

#### 12.8.1.2. Outline

The population PK analysis will be performed in the following sequence of steps:

- 1. Exploratory data analysis/data check out.
- 2. Base structural model development.
- 3. Covariate analysis.
- 4. Model refinement.
- 5. Model evaluation.
- 6. Model application using simulation

The above analysis and reporting steps follow EMEA

(http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2009/09/WC500003067.pdf) and FDA population PK guidances

(https://www.fda.gov/downloads/drugs/guidances/UCM072137.pdf)

Key components of these regulatory guidelines on population PK are also included in the Global CPMS guidance for pop pk RAP

https://connect.gsk.com/sites/cpms/TandD/Guidances

The analyses described above will be the responsibility of CPMS and will be independent of SAC. Further details will be provided in a separate RAP.

### 12.8.2. Population Pharmacokinetic (PopPK) Dataset Specification

### 12.8.2.1. Data Specification

#### 12.8.2.2. Dataset Variable Conventions

Column headings in NONMEM-ready datasets and specifications should be consistent to minimise the programming process, and facilitate a smooth transfer of projects between users as needed. IDSL standards will be followed where possible.

A list of most common standardised variable names for NONMEM datasets can be found in Table below.

File to be produced for Analyte=GSK2798745 only.

### List of Variable Names for NONMEM-Ready Datasets for PopPK Analysis

| Variable | Label (Variable description) |
|---|---|
| С | NONMEM line exclusion identifier |
| ID | NONMEM subject identifier |
| STUD | Study ID |
| SUBJID | Subject identifier for study |
| SITEID | Unique identifier for a study site |
| AMT | NONMEM Amount of drug administered then EVID =1- dose event record |
| UAMT | Unit of AMT (mg) |
| ADDL | NONMEM Additional dose |
| CONC | Drug Concentration |
| UCONC | Unit of CONC (ng/mL) |
| LNCONC | Natural log of CONC column |
| ANALYTE | Drug label e.g 745 |
| LLQ | Lower Limit of quantification |
| LNLLQ | Natural log of LLQ column |
| DAY | Study day number of record or of dosing |
| TIME<br>UTIME | Plasma sample time after last dose (actual time) Unit of TIME (h) |
| | Dose amount |
| DOSE<br>EVID | NONMEM Event ID If row has dose then EVID=1 else EVID=0 |
| EVID | If EVID=1 then this is a dose event record |
| | If $EVID = 0$ then this is an observation record |
| II | NONMEM Inter-dose interval II=24 – dose every day |
| MDV | NONMEM Missing data value then MDV=1 else MDV=0 |
| AGE | Subject Age (yrs) |
| SEX | Subject gender 0 = Male 1 = Female |
| SEXTEXT | Subject gender text Male or Female |
| BMI | Baseline Body Mass Index |
| WT | Baseline Subject weight |
| CONMED1* | Identifier for inhibitor CYP3A4 1 =Yes, 0 = No |
| CONMED1TXT* | Inhibitor Name |
| CONMED2* | Identifier for inducer CYP3A4 1 =Yes, 0 = No |
| CONMED2TXT* | Inducer Name |
| CONMED3* | Identifier for co-admin of ANY statin 1 =Yes, 0 = No |
| CONMED3TXT* | Statin name |
| CONMED4* | Identifier for co-admin of Atorvastatin 1 =Yes, 0 = No |
| CONMED4TXT* | ATORVASTATIN |
| TC 1 | rd a g CONIC has "NA" or "NS" than assign CONIC call as "" |

If observation record e.g CONC has "NA" or "NS" then assign CONC cell as "." If observation record e.g CONC has "NQ" or "BQL" then assign CONC cell as "." and MDV = 1 -this means value can be estimated by model Missing covariate data should be imputed as "-99.

Statistics & Programming in discussion with CPMS to provide dataset as specified in Table below based on column variables described above. Fields marked with a '\*' above will need discussion between S&P and CPMS prior to generating the dataset, to identify concomitant medication data applicable to each column.

| c | ID | STUD | SUBJID | SITEID | DAY | TIME | UTIME | AMT | UAMT | ADDL | II | CONC | UCONC | LNCONC | ANALYTE | LLQ | LNLLQ | MDV | EVID | AGE | WT | вмі | SEX | SEXTEXT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | PP | 207702 | PPD | | 1 | 0 | h | 4.8 | mg | 0 | 24 | | ng/mL | | 745 | 5 | 1.6 | 1 | 1 | 50 | 70 | 24 | 0 | M |
| | D | 207702 | | | 1 | 0 | h | | | 0 | | | ng/mL | | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 1 | 0.5 | h | | | 0 | | 10 | ng/mL | 2.30 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 1 | 1 | h | | | 0 | | 50 | ng/mL | 3.91 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 1 | 1.5 | h | | | 0 | | 150 | ng/mL | 5.01 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 1 | 2 | h | | | 0 | | 200 | ng/mL | 5.30 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 1 | 3.5 | h | | | 0 | | 175 | ng/mL | 5.16 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 7 | 0 | h | 2.4 | mg | 6 | 24 | | ng/mL | | 745 | 5 | 1.6 | 1 | 1 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 7 | 0.5 | h | | | 0 | | 10 | ng/mL | 2.30 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 7 | 1 | h | | | 0 | | 50 | ng/mL | 3.91 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 7 | 1.5 | h | | | 0 | | 150 | ng/mL | 5.01 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 7 | 2 | h | | | 0 | | 200 | ng/mL | 5.30 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 7 | 3.5 | h | | | 0 | | 175 | ng/mL | 5.16 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |
| | | 207702 | | | 7 | 24 | h | | | 0 | | 175 | ng/mL | 5.16 | 745 | 5 | 1.6 | 0 | 0 | 50 | 70 | 24 | 0 | M |

| CONMED1 | CONMED1TXT | CONMED2 | CONMED2TXT | CONMED3 | CONMED3TXT | CONMED4 | CONMED4TXT |
|---|---|---|---|---|---|---|---|
| 1 | INH | 0 | INDU | 1 | STATIN | 1 | ATORVASTATIN |

Notes: TIME will be actual time from dose. File to be produced just for GSK2798745. In example, CONMED3 represents 1 for a subject taking ANY statin and CONMED4 is applicable to just atorvastatin.

### 12.9. Appendix 9: Pharmacokinetic / Pharmacodynamic Analyses

### 12.9.1. Pharmacokinetic / Pharmacodynamic Methodology

### 12.9.1.1. Exposure-Response Relationship

Graphical exploration of individual predicted steady state PK exposure metric versus cough response (10-hour daily awake cough) on day 7 will be undertaken using both placebo and treatment groups. PK exposure metric for placebo group will be assigned a value of 0. If there is evidence of any trend, various PK-PD models will be explored including linear, Emax, sigmoidal Emax relationships.

PK exposure metrics include: Day 7 Cmax (predicted), Cav (predicted) and C24 (observed) on day 8

Clinical endpoint: Baseline: Day -1 & Day 7 total day-time cough count (10 hours)

Using Monte-Carlo simulations, the optimal PK-PD model for cough count will be applied to provide estimate of systemic exposure range associated with significant clinical response (10h awake cough count) from which optimal dose of GSK2798745 can be estimated for future studies, taking into account estimate of PK variability of parent drug.

The analyses described above will be the responsibility of CPMS and will be independent of SAC. Further details will be provided in a separate RAP.

### 12.9.2. Pharmacokinetic / Pharmacodynamic Dataset Specification

### 12.9.2.1. Data Specification

#### 12.9.2.2. Dataset Variable Conventions

Column headings in NONMEM-ready datasets and specifications should be consistent to minimise the programming process, and facilitate a smooth transfer of projects between users as needed. IDSL standards will be followed where possible.

A list of most common standardised variable names for NONMEM datasets can be found in Table below

File to be produced for Analyte=GSK2798745 only.

#### List of Variable Names for NONMEM-Ready Datasets for Pop PK-PD Analysis

| Variable | Label (Variable description) | Source (other sources may |
|----------|----------------------------------|-------------------------------|
| | | be used) |
| С | NONMEM line exclusion identifier | Derived as '.' – see example, |
| | | required for software |
| ID | NONMEM subject identifier | Derived – set to PPD etc & |
| | | linked to SUBJID – see |
| | | example |
| STUD | Study ID | ARDATA.POP (STUDYID) |

| Variable | Label (Variable description) | Source (other sources may be used) |
|---|---|---|
| SUBJID | Subject identifier for study | ARDATA.POP (SUBJID) |
| SITEID | Unique identifier for a study site | ARDATA.POP |
| | | (CENTREID) |
| DAY | Study day Day -1 10h cough count before dosing. | PKCNC (derive from VISIT) |
| DIZ 1 | Day 7 10h cough count after day 7 dose | |
| PK1 | Predicted Cmax on day 7 – Provided by POPPK analysis* | Create variable but leave blank |
| PK2 | Predicted Cav on day 7 - Provided by POPPK | Create variable but leave |
| 1112 | analysis* | blank |
| PK3 | Predicted C24 on day 8 - Provided by POPPK | Create variable but leave |
| | analysis* | blank |
| Analyte | GSK2798745 | ARDATA.PKCNC |
| R10BASE1 | Raw baseline 10h cough count before period 1 | ARDATA.COUGHTOT (see |
| R10BASE2 | Raw baseline 10h cough count before period 2 | notes) As above |
| RPD10 | Raw 10h awake cough count [primary endpoint] | As above |
| R24BASE1 | Raw baseline 24h cough count before period 1 | As above |
| R24BASE2 | Raw baseline 24h cough count before period 2 | As above |
| RPD24 | Raw 24h cough count total | As above |
| I10BASE1 | Imputed baseline 10h cough count before period 1 | As above |
| I10BASE2 | Imputed baseline 10h cough count before period 2 | As above |
| IPD10 | Imputed 10h awake cough count [primary endpoint] | As above |
| I24BASE1 | Imputed baseline 24h cough count before period 1 | As above |
| I24BASE2 | Imputed baseline 24h cough count before period 2 | As above |
| IPD24 | Imputed 24h cough count total | As above |
| F10BASE1 | Flag for imputed baseline 10h cough count before period 1 | As above |
| F10BASE2 | Flag for imputed baseline 10h cough count before period 2 | As above |
| FPD10 | Flag for imputed 10h awake cough count [primary endpoint] | As above |
| F24BASE1 | Flag for imputed baseline 24h cough count before period 1 | As above |
| F24BASE2 | Flag for imputed baseline 24h cough count before period 2 | As above |
| FPD24 | Flag for imputed 24h cough count total | As above |
| AGE | Subject Age (yrs) | ARDATA.DEMO |
| SEX | Subject gender 0 = Male 1 = Female | ARDATA.DEMO |
| SEXTEXT | Subject gender text Male or Female | ARDATA.DEMO |
| BMI | Baseline Body Mass Index | ARDATA.DEMO |
| WT | Baseline Subject weight | ARDATA.DEMO |
| TMT | 1 = Placebo ; 2 = Drug | ARDATA.TRT |
| TMTTEXT | Treatment text Placebo or GSK2798745 | ARDATA.TRT |

| Variable | Label (Variable description) | Source (other sources may be used) |
|---|---|---|
| PERIOD | 1 = Period 1; $2 = Period 2$ | ARDATA.TRT |

Statistics & Programming in discussion with CPMS to provide dataset as specified in Table below based on column variables described above.

\*The predicted POPPK parameters detailed above will be generated by CPMS. The Pop PK-PD dataset above will be generated by programming with these variables included as blank, for CPMS to populate at a later date.

### Note to programmers for cough data:

Variables, R\*, I\* and F\* can be obtained from A&R dataset COUGHTOT. Cough totals are COUGHTOT (raw totals) and COUGHIMP (imputed totals) Select where FLAGHR=100 and FLAGHR=240 to get 10h and 24h totals. Select where VISITNUM in (20, 60) to get Day -1 totals for Period 1 and 2. Select where VISITNUM in (40, 80) to get Day 7 totals for Period 1 and 2. FLAGIMP will indicate if imputation occurred at timepoint of interest.

# 

| С | D STUE | SIT | EID SUBJII | DAY | PK1 | PK2 | PK3 | ANALYTE | R10BASE1 | R10BASE2 | RPD10 | R24BASE1 | R24BASE2 | RPD24 | I10BASE1 | I10BASE2 | IPD10 | I24BASE1 | I24BASE2 | IPD24 | AGE | WT | BMI | SEX | SEXTXT | TMT | TMTTEXT | PERIOD |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ļ. F | P 2077 | 702 I | PPD | -1 | l | | | GSK2798745 | 25 | 23 | 25 | 80 | 75 | 80 | 25 | 23 | 25 | 80 | 75 | 80 | 50 | 70 | 24 | 0 | M | 1 | Placebo | 1 |
| | 2077 | 702 | | 7 | 7 | | | GSK2798745 | 25 | 23 | 23 | 80 | 75 | 60 | 25 | 23 | 23 | 80 | 75 | 60 | 50 | 70 | 24 | 0 | M | 1 | Placebo | 1 |
| | 2077 | 702 | | -1 | l | | | GSK2798745 | 25 | 23 | 23 | 80 | 75 | 75 | 25 | 23 | 23 | 80 | 75 | 75 | 50 | 70 | 24 | 0 | M | 2 | GSK2798745 | 2 |
| | 2077 | 702 | | 7 | 7 | | | GSK2798745 | 25 | 23 | 10 | 80 | 75 | 55 | 25 | 23 | 10 | 80 | 75 | 60 | 50 | 70 | 24 | 0 | M | 2 | GSK2798745 | 2 |
| | 2077 | 702 | | -1 | | | | GSK2798745 | 30 | 28 | 30 | 55 | 57 | 55 | 30 | 28 | 30 | 55 | 57 | 55 | 60 | 75 | 24 | 1 | F | 2 | GSK2798745 | 1 |
| | 2077 | 702 | | 7 | 7 | | | GSK2798745 | 30 | 28 | 12 | 55 | 57 | 40 | 30 | 28 | 12 | 55 | 57 | 40 | 60 | 75 | 24 | 1 | F | 2 | GSK2798745 | 1 |
| | 2077 | 702 | | -1 | | | | GSK2798745 | 30 | 28 | 28 | 55 | 57 | 57 | 30 | 28 | 28 | 55 | 57 | 57 | 60 | 75 | 24 | 1 | F | 1 | Placebo | 2 |
| | 2077 | 702 | | 7 | 7 | | | GSK2798745 | 30 | 28 | 25 | 55 | 57 | 50 | 30 | 28 | 25 | 55 | 57 | 60 | 60 | 75 | 24 | 1 | F | 1 | Placebo | 2 |

# 12.10. Appendix 10: Abbreviations & Trade Marks

### 12.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| ALT | Alanine aminotranferase |
| A&R | Analysis and Reporting |
| AST | Aspartate aminotransferase |
| AUC | Area under the concentration time curve |
| BMI | Body mass index |
| BUN | Blood urea nitrogen |
| Cav | Average concentration of drug over the dosing interval |
| CI | Confidence Interval |
| Cmax | Maximum observed plasma concentration |
| CPK | Creatinine phosphokinase |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CPSR | Clinical Pharmacology Study Report |
| CSSRS | Columbia Suicidality Severity Rating Scale |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FOBT | Faecal Occult Blood Test |
| GSK | GlaxoSmithKline |
| h | Hours |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| LCQ | Leicester Cough Questionnaire |
| LDH | Lactate dehydrogenase |
| LLN | Lower limit of normal |
| MCH | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular volume |
| mg | Milligrams |
| MHRA | Medicine and Healthcare Products Regulatory Agency |
| mm | Millimetres |
| MMRM | Mixed Model Repeated Measures |
| N | Number |

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RBC | Red blood cells |
| S&P | Statistics and Programming |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event(s) |
| SI | System Independent |
| SOP | Standard Operation Procedure |
| TFL | Tables, Figures & Listings |
| Tmax | Time to maximum observed concentration |
| UK | United Kingdom |
| ULN | Upper limit of normal |
| VAS | Visual Analogue Scale |
| WBC | White blood cells |

### 12.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| HARP |
| RANDALL NG |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| WinNonlin |
| SAS |
| NONMEM |

### 12.11. Appendix 11: List of Data Displays

### 12.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Population Pharmacokinetic (PopPK) | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacodynamic and / or Biomarker | 6.1 to 6.n | 6.1 to 6.n |
| Pharmacokinetic / Pharmacodynamic | 7.1 to 7.n | 7.1 to 7.n |
| Section | List | ings |
| ICH Listings | 1 t | 0 X |
| Other Listings | y to z | |

Note that all displays (Tables, Figures & Listings) will use the term 'Subjects'.

### 12.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|----------|----------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Population Pharmacokinetic (PopPK) | POPPK_Fn | POPPK_Tn | POPPK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 12.11.3. Deliverables

| Delivery [Priority] [1] | Description |
|---|---|
| IA GSK [X] | Interim Analysis Statistical Analysis Complete – Outputs to be generated by GSK |
| SAC [X] | SAC [X] Final Statistical Analysis Complete – Outputs to be generated by FSP |
| SAC GSK [X] | Final Statistical Analysis Complete – Outputs to be generated by <b>GSK</b> |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 12.11.4. Study Population Tables

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Subject Disposition | | | | |
| 1.1. | All Subjects | ES1A | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC [2] |
| 1.2. | All Subjects | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC [2] |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC [2] |
| Protoco | Protocol Deviation | | | | |
| 1.4. | All Subjects | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC [2] |
| Popula | Population Analysed | | | | |
| 1.5. | All Subjects | SP1A | Summary of Study Populations | IDSL | SAC [2] |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1.6. | All Subjects | DM3 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC [2] |
| 1.7. | All Subjects | DM11 | Summary of Age Ranges | EudraCT | SAC [2] |
| 1.8. | All Subjects | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC [2] |
| Prior ar | Prior and Concomitant Medications | | | | |
| 1.9. | All Subjects | MH1 | Summary of Past Medical Conditions | ICH E3 | SAC [2] |
| 1.10. | All Subjects | MH1 | Summary of Current Medical Conditions | ICH E3 | SAC [2] |
| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.11. | All Subjects | CM1 | Summary of Concomitant Medications | ICH E3 See IDSL for options related to ATC groupings and multi-ingredient medications. | SAC [2] |
| Exposu | re and Treatmen | t Compliance | | | |
| 1.12. | All Subjects | EX1 | Summary of Exposure to Study Treatment | ICH E3 Dose and/or time on treatment, as applicable. Many possible considerations; defer to therapy area standards where available. | SAC [2] |
| 1.13. | All Subjects | POP_L1 | Listing of Compliance | | SAC [2] |

### 12.11.5. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 10H To | tal Cough Cour | nt | | | |
| 2.1. | All Subjects | EF_T2 | Summary of Day-Time 10h Total Cough Counts | Include raw cough counts and imputed cough counts as per mock-up, geometric means for log-transformed data on second page | SAC GSK [1] |
| 2.2. | All Subjects | EF_T1 | Summary of Statistical Analysis of Day-Time 10h Total Cough Counts at Day 7 | Statistical analysis to be based on imputed cough counts | IA GSK, SAC<br>GSK [1] |
| 2.3. | All Subjects | EF_T1 | Summary of Statistical Analysis of Day-Time 10h Total Cough Counts at Day 7 (Sensitivity) | Statistical analysis to be based on <b>non-imputed</b> cough counts | SAC GSK [1] |
| 24H To | tal Cough Cour | nt | | | |
| 2.4. | All Subjects | EF_T2 | Summary of 24h Total Cough Counts | Include raw cough counts and imputed cough counts as per mock-up, geometric means for log-transformed data on second page | SAC GSK [1] |
| 2.5. | All Subjects | EF_T1 | Summary of Statistical Analysis of 24h Total Cough Counts at Day 7 | Statistical analysis to be based on imputed cough counts | SAC GSK [1] |
| 2.6. | All Subjects | EF_T1 | Summary of Statistical Analysis of 24h Total Cough Counts atDay 7 (Sensitivity) | Statistical analysis to be based on <b>non-imputed</b> cough counts | SAC GSK [1] |
| Severit | y of Cough (VA | S) | | , | |
| 2.7. | All Subjects | EF_T3 | Summary of Severity of Cough (VAS) | Collected at Screening, D1(Pre-Dose), D7(Pre-Dose) and FU | SAC [2] |
| 2.8. | All Subjects | EF_T4 | Summary of Change From Baseline in Severity of Cough (VAS) | Include change from baseline to D7(Pre-Dose) only | SAC [2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.9. | All Subjects | EF_T5 | Summary of Statistical Analysis of Change From Baseline in Severity of Cough (VAS) at Day 7 | Analysis of change from baseline D1(Pre-Dose) to D7(Pre-Dose) | SAC [2] |
| Urge to | Cough (VAS) | | | | |
| 2.10. | All Subjects | EF_T3 | Summary of Urge to Cough (VAS) | Collected at D1(Pre-Dose), D7(Pre-<br>Dose) and FU | SAC [2] |
| 2.11. | All Subjects | EF_T4 | Summary of Change From Baseline in Urge to Cough (VAS) | Include change from baseline to D7(Pre-Dose) only | SAC [2] |
| 2.12. | All Subjects | EF_T5 | Summary of Statistical Analysis of Change From Baseline in Urge to Cough (VAS) at Day 7 | Analysis of change from baseline D1(Pre-Dose) to D7(Pre-Dose) | SAC [2] |
| Leicest | ter Cough Ques | stionnaire (LCQ) | | | |
| 2.13. | All Subjects | EF_T6 | Summary of the Leicester Cough Questionnaire (LCQ) | Summarise each of the 3 domains and an overall total score. Collected at D1(Pre-Dose) and D7(Pre-Dose) | SAC [2] |
| 2.14. | All Subjects | EF_T7 | Summary of Change From Baseline in the Leicester Cough Questionnaire (LCQ) | Include change from baseline to D7(Pre-Dose) for domain scores and total | SAC [2] |
| 2.15. | All Subjects | EF_T8 | Statistical Analysis of Change From Baseline in the Leicester Cough Questionnaire (LCQ) at Day 7 | 4 x analyses, one for each domain and overall score | SAC [2] |

### 12.11.6. Efficacy Figures

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 10H To | tal Cough Cou | nt and 24 Total Co | ugh Count | | |
| 2.1. | All Subjects | EF_F1 | Summary of Geometric Means and 95% CI for Baseline and Day 7 10h Day-time Cough Counts, by Treatment Group | Footnote to include 'Note: Imputed data is presented, where cough counts are pro-rated based on a minimum of 60% of data being available' | IA GSK, SAC<br>GSK [1] |
| 2.2. | All Subjects | EF_F1 | Summary of Geometric Means and 95% CI for Baseline and Day 7 24h Day-time Cough Counts, by Treatment Group | Follow example EF_F1 but use 24 hour totals (imputed). Footnote as above. | SAC GSK [1] |
| 2.3. | All Subjects | EF_F2 | Summary of Geometric Means and 95% CI by Hourly Intervals (0-10h) for Day 7 Cough Counts | If zero counts are present and log-<br>transformation of hourly totals not<br>possible, then this figure will present<br>arithmetic means and 95% CI instead.<br>Footnote as above. | IA GSK, SAC<br>GSK [1] |
| 2.4. | All Subjects | EF_F2 | Summary of Geometric Means and 95% CI by Hourly Intervals (0-24h) for Day 7 Cough Counts | If zero counts are present and log-<br>transformation of hourly totals not<br>possible, then this figure will present<br>arithmetic means and 95% CI instead.<br>Footnote as above. | SAC GSK [1] |
| 2.5. | All Subjects | EF_F3 | Individual Subject Profiles of Cough Count Totals by 1 Hour Intervals (0-10h) Day 7 | 4 subjects per page, hourly timepoint e.g 0-1h, 1-2h etc on the x-axis, cough total on the y-axis, treatment group in a legend. Display imputed hourly data (pro-rated) for this plot. Footnote as above. | SAC GSK [1] |

| Efficac | y: Figures | IDSL / | | | Dalivarahla |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.6. | All Subjects | EF_F3 | Individual Subject Profiles of Cough Count Totals by 1 Hour Intervals (0-24h) Day 7 | 4 subjects per page, hourly timepoint e.g 0-1h, 1-2h etc on the x-axis, cough total on the y-axis, treatment group in a legend. Extend to 24h. Display imputed hourly data (pro-rated) for this plot. Footnote as above. | SAC GSK [1] |
| 2.7. | All Subjects | EF_F4 | Boxplots of Cough Count Totals by 1 Hour Intervals (0-10h) Day 7 | Hourly timepoint e.g 0-1h, 1-2h etc on the x-axis. Cough count total on the y-axis. Treatment group in a legend. Display imputed hourly data (pro-rated) for this plot. Footnote as above. | SAC GSK [1] |
| 2.8. | All Subjects | EF_F4 | Boxplots of Cough Count Totals by 1 Hour Intervals (0-24h) Day 7 | Hourly timepoint e.g 0-1h, 1-2h etc on the x-axis. Cough count total on the y-axis. Treatment group in a legend. Display imputed hourly data (pro-rated) for this plot. Extend to 24h. Footnote as above. | SAC GSK [1] |
| 2.9. | All Subjects | EF_F5 | Individual 10h Cough Counts Day 7 | Subject on the x-axis and 10h totals by treatment on the y-axis, with a legend for treatment group. Display imputed 10h data (pro-rated). Footnote as above. | SAC GSK [1] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10. | All Subjects | EF_F5 | Individual 24h Cough Counts Day 7 | Subject on the x-axis and 24h totals by treatment on the y-axis, with a legend for treatment group. Display imputed 24h data (pro-rated). Follow example EF_F5 but extend to 24h. Footnote as above. | SAC GSK [1] |
| 2.11. | All Subjects | EF_F6 | Individual Changes From Baseline in 10h Day-time Cough<br>Counts | Individual subjects changes from baseline (Day -1) to Day 7 by treatment. 10h totals. Footnote as above. | SAC GSK [1] |
| 2.12. | All Subjects | EF_F6 | Individual Changes From Baseline in 24h Day-time Cough<br>Counts | Individual subjects changes from baseline (Day -1) to Day 7 by treatment. 24h totals. Footnote as above. | SAC GSK [1] |
| 2.13. | All Subjects | EF_F7 | Adjusted Median Responses and 95% Cr. Intervals for 10h Total Cough Counts on Day 7 | X-axis can say 'Day 7'. Y-axis will be median cough counts with 95% Crls (back-transformed estimates). Treatment group in a legend. Footnote as per mock example. | SAC GSK [1] |
| 2.14. | All Subjects | EF_F7 | Adjusted Median Responses and 95% Cr. Intervals for 24h Total Cough Counts on Day 7 | X-axis can say 'Day 7'. Y-axis will be median cough counts and 95% Crls (back-transformed estimates). Treatment group in a legend. Footnote as per mock example. | SAC GSK [1] |
| 2.15. | All Subjects | EF_F1 | Summary of Geometric Means and 95% CI for Baseline and Day 7 10h Day-time Cough Counts, by Treatment Group by Prior Cough Study Participation | Footnote to include 'Note: Imputed data is presented, where cough counts are pro-rated based on a minimum of 60% of data being available' | SAC GSK [2] |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.16. | All Subjects | EF_F1 | Summary of Geometric Means and 95% CI for Baseline and Day 7 24h Day-time Cough Counts, by Treatment Group by Prior Cough Study Participation | Follow example EF_F1 but use 24 hour totals (imputed). Footnote as above. | SAC GSK [2] |
| 2.17. | All Subjects | EF_F2 | Summary of Geometric Means and 95% CI by Hourly Intervals (0-10h) for Day 7 Cough Counts by Prior Cough Study Participation | If zero counts are present and log-<br>transformation of hourly totals not<br>possible, then this figure will present<br>arithmetic means and 95% CI instead.<br>Footnote as above. | SAC GSK [2] |
| 2.18. | All Subjects | EF_F2 | Summary of Geometric Means and 95% CI by Hourly Intervals (0-24h) for Day 7Cough Counts by Prior Cough Study Participation | If zero counts are present and log-<br>transformation of hourly totals not<br>possible, then this figure will present<br>arithmetic means and 95% CI instead.<br>Footnote as above. | SAC GSK [2] |
| 2.19. | All Subjects | EF_F6 | Individual Changes From Baseline in 10h Day-time Cough<br>Counts by Period | Individual subjects changes from baseline (Day -1) to Day 7 by treatment and period. 10h totals. Footnote as above. | SAC GSK [1] |
| 2.20. | All Subjects | EF_F6 | Individual Changes From Baseline in 24h Day-time Cough<br>Counts by Period | Individual subjects changes from baseline (Day -1) to Day 7 by treatment and period. 24h totals. Footnote as above. | SAC GSK [1] |
| 2.21. | All Subjects | EF_F1 | Summary of Geometric Means and 95% CI for Baseline and Day 7 10h Day-time Cough Counts, by Treatment Group and Period | Footnote as above. | IA GSK, SAC<br>GSK [1] |
| 2.22. | All Subjects | EF_F1 | Summary of Geometric Means and 95% CI for Baseline and Day 7 24h Day-time Cough Counts, by Treatment Group and Period | Footnote as above. | SAC GSK [1] |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Severit | y of Cough (VA | iS) | | | |
| 2.23. | All Subjects | EF_F1 | Summary of Severity of Cough (VAS) (Means $\pm$ 95% CI) by Visit | X-axis will be Day -1 and Day 7. Y-axis will be mean cough severity $\pm$ 95% CI. Similar to example EF_F1 but with arithmetic means. | SAC [2] |
| 2.24. | All Subjects | EF_F7 | Adjusted Median Responses and 95% Cr. Intervals for Change From Baseline in Severity of Cough (VAS) | X-axis can say 'Day 7 (PD)'. Y-axis will be median CFB cough severity and 95% Crls. Treatment group in a legend or on x-axis. | SAC [2] |
| Urge to | Cough (VAS) | | | | |
| 2.25. | All Subjects | EF_F1 | Summary of Urge to Cough (VAS) (Means $\pm$ 95% CI) by Visit | X-axis will be Day -1 and Day 7. Y-axis will be mean urge to cough ± 95% CI. Similar to example EF_F1 but with arithmetic means. | SAC [2] |
| 2.26. | All Subjects | EF_F7 | Adjusted Median Responses and 95% Cr. Intervals for Change From Baseline in Urge to Cough (VAS) | X-axis can say 'Day 7 (PD)'. Y-axis will be median CFB urge to cough and 95% Crls. Treatment group in a legend or on x-axis. | SAC [2] |
| Leicest | ter Cough Ques | stionnaire (LCQ) | | | |
| 2.27. | All Subjects | EF_F1 | Summary of Leicester Cough Questionnaire (LCQ) (Means $\pm$ 95% CI) by Visit | X-axis will be Day -1 and Day 7. Y-axis will be mean score ± 95% CI. 4 pages one for each of the 3 domains and one for total score. | SAC [2] |
| | | | | Similar to example EF_F1 but with arithmetic means. | |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.28. | All Subjects | EF_F7 | Adjusted Median Responses and 95% Cr. Intervals for Change From Baseline in Leicester Cough Questionniare (LCQ) | X-axis can say 'Day 7 (PD)'. Y-axis will be median CFB LCQ score and 95% Crls. Treatment group in a legend or on x-axis. 4 pages one for each of the 3 domains and one for total score | SAC [2] |

# 12.11.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | All Subjects | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC [2] |
| 3.2. | All Subjects | AE1CP | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term/by Overall Frequency | ICH E3 | SAC [2] |
| Serious | and Other Sig | nificant Adverse I | Events | | |
| 3.3. | All Subjects | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC [2] |
| Laborat | Laboratory: Chemistry | | | | |
| 3.4. | All Subjects | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | SAC [2] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Hematolo | gy | | | |
| 3.5. | All Subjects | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC [2] |
| ECG | | | | | |
| 3.6. | All Subjects | EG1 | Summary of ECG Findings | IDSL | SAC [2] |
| 3.7. | All Subjects | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC [2] |
| Vital Si | gns | | | | |
| 3.8. | All Subjects | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3<br>Include Weight as well as Blood<br>Pressure, HR and Temperature | SAC [2] |
| CSSRS | | I | | | |
| 3.9. | All Subjects | CSSRS4 | Listing of C-SSRS Suicidal Ideation and Behaviour Data | Refer to IDSL guidance and example CSSRS4. For studies with very few suicical events expected, this listing can substitute the summary table. | SAC [2] |
| Audion | netry | | | | |
| 3.10. | All Subjects | SAF_L1 | Listing of Audiometry | Add footnote: Pre-Treatment Period 1 audiometry can be done anytime between Screening and Treatment Period 1, Day 1, pre-dose. Pre-Treatment Period 2 audiometry can be done any time during the washout period (up to Treatment Period 2, Day 1 pre-dose). | SAC [2] |

### 12.11.8. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | centration | | | | |
| 4.1. | PK | PKCT1 (PK01) | Summary of <b>GSK2798745</b> Pharmacokinetic Concentration-Time Data (ng/mL) | | SAC [2] |
| 4.2. | PK | PKCT1 (PK01) | Summary of <b>GSK2798745 M1 Metabolite</b> Pharmacokinetic Concentration-Time Data (ng/mL) | | SAC [2] |
| 4.3. | PK | PKCT1 (PK01) | Summary of <b>Atorvastatin</b> Pharmacokinetic Concentration-Time Data (ng/mL) | Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |
| 4.4. | PK | PKCT1 (PK01) | Summary of <b>Atorvastatin Metabolite</b> Pharmacokinetic Concentration-Time Data (ng/mL) | Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Par | ameter | | | | |
| 4.5. | PK | PKPT1 (PK03) | Summary Statistics of Derived Plasma <b>GSK2798745</b> Pharmacokinetic Parameters | | SAC [2] |
| 4.6. | PK | PKPT1 (PK03) | Summary Statistics of Derived Plasma GSK2798745 M1 Metabolite Pharmacokinetic Parameters | | SAC [2] |
| 4.7. | PK | PKPT1 (PK03) | Summary Statistics of Derived Plasma <b>Atorvastatin</b> Pharmacokinetic Parameters | | SAC [2] |
| 4.8. | PK | PKPT1 (PK03) | Summary Statistics of Derived Plasma <b>Atorvastatin Metabolite</b> Pharmacokinetic Parameters | | SAC [2] |
| 4.9. | PK | PKPT3 (PK05) | Summary Statistics of Log-Transformed Derived Plasma GSK2798745 Pharmacokinetic Parameters | | SAC [2] |
| 4.10. | PK | PKPT3 (PK05) | Summary Statistics of Log-Transformed Derived Plasma GSK2798745 M1 Metabolite Pharmacokinetic Parameters | | SAC [2] |
| 4.11. | PK | PKPT3 (PK05) | Summary Statistics of Log-Transformed Derived Plasma Atorvastatin Pharmacokinetic Parameters | | SAC [2] |
| 4.12. | PK | PKPT3 (PK05) | Summary Statistics of Log-Transformed Derived Plasma Atorvastatin Metabolite Pharmacokinetic Parameters | | SAC [2] |

# 12.11.9. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 4.1. | PK | PKCF1X<br>(PK16b) | Individual <b>GSK2798745</b> Plasma Concentration—Time Plots (Linear and Semi-log) | By Subject plots – by visit (Day 1 pre-dose to 3.5h profile and Day 7 pre-dose to 24h profile) | SAC [2] |
| 4.2. | PK | PKCF6 (PK24) | Individual <b>GSK2798745</b> Plasma Concentration—Time Plot (Linear and Semi-log) | Limit to 12 subjects per graphic split over pages (e.g. 2 pages for N=24, 3 pages for N=36) | SAC [2] |
| 4.3. | PK | PKCF2 (PK17) | Mean Plasma <b>GSK2798745</b> Concentration-Time Plot (Linear and Semi-Log) | | SAC [2] |
| 4.4. | PK | PKCF3 (PK18) | Median Plasma <b>GSK2798745</b> Concentration-Time Plot (Linear and Semi-Log) | | SAC [2] |
| 4.5. | PK | PKCF1X<br>(PK16b) | Individual <b>GSK2798745 Metabolite M1</b> Plasma Concentration—<br>Time Plots (Linear and Semi-log) | By Subject plots – by visit (Day 1 pre-dose to 3.5h profile and Day 7 pre-dose to 24h profile) | SAC [2] |
| 4.6. | PK | PKCF6 (PK24) | Individual <b>GSK2798745 Metabolite M1</b> Plasma Concentration—<br>Time Plot<br>(Linear and Semi-log) | Limit to 12 subjects per graphic split over pages (e.g. 2 pages for N=24, 3 pages for N=36) | SAC [2] |

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.7. | PK | PKCF2 (PK17) | Mean Plasma <b>GSK2798745 Metabolite M1</b> Concentration-Time Plot (Linear and Semi-Log) | | SAC [2] |
| 4.8. | PK | PKCF3 (PK18) | Median Plasma <b>GSK2798745 Metabolite M1</b> Concentration-<br>Time Plot (Linear and Semi-Log) | | SAC [2] |
| 4.9. | PK | PKCF1X<br>(PK16b) | Individual <b>Atorvastatin</b> Plasma Concentration–Time Plots (Linear and Semi-log) | By Subject plots – by visit (Day 1 pre-dose to 3.5h profile and Day 7 pre-dose to 24h profile) Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |
| 4.10. | PK | PKCF6 (PK24) | Individual <b>Atorvastatin</b> Plasma Concentration–Time Plot (Linear and Semi-log) | Limit to 12 subjects per graphic split over pages (e.g. 2 pages for N=24, 3 pages for N=36) Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |
| 4.11. | PK | PKCF2 (PK17) | Mean Plasma <b>Atorvastatin</b> Concentration-Time Plot (Linear and Semi-Log) | Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |
| 4.12. | PK | PKCF3 (PK18) | Median Plasma <b>Atorvastatin</b> Concentration-Time Plot (Linear and Semi-Log) | Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.13. | PK | PKCF1X<br>(PK16b) | Individual <b>Atorvastatin Metabolite</b> Plasma Concentration–Time Plots (Linear and Semi-log) | By Subject plots – by visit (Day 1 pre-dose to 3.5h profile and Day 7 pre-dose to 24h profile) Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |
| 4.14. | PK | PKCF6 (PK24) | Individual <b>Atorvastatin Metabolite</b> Plasma Concentration–Time Plot (Linear and Semi-log) | Limit to 12 subjects per graphic split over pages (e.g. 2 pages for N=24, 3 pages for N=36) Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |
| 4.15. | PK | PKCF2 (PK17) | Mean Plasma <b>Atorvastatin Metabolite</b> Concentration-Time Plot (Linear and Semi-Log) | Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |
| 4.16. | PK | PKCF3 (PK18) | Median Plasma <b>Atorvastatin Metabolite</b> Concentration-Time Plot (Linear and Semi-Log) | Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |

# 12.11.10. ICH Listings

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC [2] |
| 2. | All Subjects | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC [2] |
| 3. | All Subjects | SD3 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC [2] |
| 4. | All Subjects | BL2 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC [2] |
| 5. | All Subjects | CP_RA1x | Listing of Planned and Actual Treatments | IDSL | SAC [2] |
| Protoc | ol Deviations | 1 | | | |
| 6. | All Subjects | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC [2] |
| 7. | All Subjects | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC [2] |
| Popula | tions Analysed | | | | 1 |
| 8. | All Subjects | SP3a | Listing of Participants Excluded from Any Population | ICH E3 | SAC [2] |
| Demog | raphic and Bas | seline Characteris | tics | | , |
| 9. | All Subjects | DM4 | Listing of Demographic Characteristics | ICH E3 | SAC [2] |
| 10. | All Subjects | DM10 | Listing of Race | ICH E3 | SAC [2] |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | All Subjects | CP_CM4 | Listing of Concomitant Medications | IDSL | SAC |
| Exposi | re and Treatme | ent Compliance | | | |
| 12. | All Subjects | EX4 | Listing of Exposure Data | ICH E3 | SAC [2] |
| Advers | e Events | | | | |
| 13. | All Subjects | AE9CP | Listing of All Adverse Events | ICH E3 | SAC [2] |
| 14. | All Subjects | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC [2] |
| Serious | s and Other Sig | nificant Adverse l | Events | | |
| 15. | All Subjects | AE9CPa | Listing of Serious Adverse Events | ICH E3 | SAC [2] |
| 16. | All Subjects | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3. Provides additional detail from SAE form e.g hospitalisation (Y/N) etc | SAC [2] |
| 17. | All Subjects | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC [2] |
| All Lab | oratory | | | | |
| 18. | All Subjects | LB6 | Listing of All Clinical Chemistry Data for Participants with Any Value of Potential Clinical Importance/Outside Normal Range | ICH E3 | SAC [2] |
| 19. | All Subjects | LB6 | Listing of Clinical Chemistry Values of Potential Clinical Importance | | SAC [2] |
| 20. | All Subjects | LB6 | Listing of All Hematology Data for Participants with Any Value of Potential Clinical Importance/Outside Normal Range | | SAC [2] |
| 21. | All Subjects | LB6 | Listing of Hematology Values of Potential Clinical Importance | | SAC [2] |
| 22. | All Subjects | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC [2] |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 23. | All Subjects | UR2B | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC [2] |
| ECGs | | | | | |
| 24. | All Subjects | EG4 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL | SAC [2] |
| 25. | All Subjects | EG4 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC [2] |
| 26. | All Subjects | EG6 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC [2] |
| 27. | All Subjects | EG6 | Listing of Abnormal ECG Findings | IDSL | SAC [2] |
| Vital Si | Vital Signs | | | | |
| 28. | All Subjects | VS5 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC [2] |
| 29. | All Subjects | VS5 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC [2] |

# 12.11.11. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 30. | All Subjects | EF_L1 | Listing of Hourly and Total Cough Counts | | SAC GSK [1] |
| 31. | All Subjects | EF_L2 | Listing of Severity and Urge to Cough (VAS) | | SAC [2] |
| 32. | All Subjects | EF_L3 | Listing of Leicester Cough Questionnaire (LCQ) | | SAC [2] |
| 33. | All Subjects | - | Listing of SAS Output for 10h Total Cough Count Analysis | | SAC GSK [1] |
| 34. | All Subjects | - | Listing of SAS Output for 24h Total Cough Count Analysis | | SAC GSK [1] |
| 35. | All Subjects | - | Listing of SAS Output for CFB Severity to Cough Analysis | | SAC [2] |
| 36. | All Subjects | - | Listing of SAS Output for CFB Urge to Cough Analysis | | SAC [2] |
| 37. | All Subjects | - | Listing of SAS Output for CFB Leicester Cough Questionnaire Analysis | | SAC [2] |
| 38. | PK | PKCL1X<br>(PK08) | Listing of <b>GSK2798745</b> Plasma Pharmacokinetic Concentration–Time Data | | SAC [2] |
| 39. | PK | PKPL1X<br>(PK14) | Listing of Derived <b>GSK2798745</b> Plasma Pharmacokinetic Parameters | | SAC [2] |
| 40. | PK | PKCL1X<br>(PK08) | Listing of <b>GSK2798745 Metabolite M1</b> Plasma Pharmacokinetic Concentration–Time Data | | SAC [2] |
| 41. | PK | PKPL1X<br>(PK14) | Listing of Derived <b>GSK2798745 Metabolite M1</b> Plasma Pharmacokinetic Parameters | | SAC [2] |
| 42. | PK | PKCL1X<br>(PK08) | Listing of <b>Atorvastatin</b> Plasma Pharmacokinetic Concentration—<br>Time Data | | SAC [2] |
| 43. | PK | PKPL1X<br>(PK14) | Listing of Derived <b>Atorvastatin</b> Plasma Pharmacokinetic Parameters | | SAC [2] |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 44. | PK | PKCL1X<br>(PK08) | Listing of <b>Atorvastatin Metabolite</b> Plasma Pharmacokinetic Concentration–Time Data | Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |
| 45. | PK | PKPL1X<br>(PK14) | Listing of Derived <b>Atorvastatin Metabolite</b> Plasma<br>Pharmacokinetic Parameters | Add footnote 'Planned Relative Time is based on last dose of GSK2798745 but the timing of the last dose of Atorvastatin may vary.' | SAC [2] |

207702

# 12.12. Appendix 12: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request